

# CONFIDENTIAL

# **Statistical Analysis Plan (SAP)**

| Sponsor: | Blue Earth Diagnostics Ltd. |
|---|---|
| Study code: | BED-PSMA-101 |
| CTC project no: | 213-22-2018 |
| Study title: | A phase I, open-label study to assess safety, biodistribution, and internal radiation dosimetry of <sup>18</sup> F-rhPSMA-7.3 injection in healthy volunteers, and to assess safety and investigate the imaging characteristics in subjects with prostate cancer. |
| SAP version and date: | 30OCT2019 – Final v 1.0 |



Protocol Version No: 190222\_BED\_CSP\_v1.0\_final

Study Code: BED-PSMA-101 CTC Project No: 213-22-2018

| 1 | VE | RSION HISTORY | 5 |
|---|-------|--------------------------------------------------|----|
| 2 | INT | TRODUCTION | 5 |
| 3 | CL | INICAL STUDY DETAILS | 6 |
| | 3.1 | Clinical Study Objectives and Endpoints | 6 |
| | 3.2 | Clinical Study Design | 7 |
| | 3.3 | Statistical Hypotheses | 7 |
| | 3.4 | Number of Subjects | 7 |
| | 3.5 | Evaluability criteria | 7 |
| | 3.6 | Methods of Assigning Subject to IMP | 8 |
| | 3.7 | Blinding | 8 |
| 4 | ST | ATISTICAL AND ANALYTICAL PLANS | 9 |
| | 4.1 | Sample Size Determination | 9 |
| | 4.2 | Definition of Analysis Sets | 9 |
| | 4.2.1 | Safety Analysis Set | 9 |
| | 4.2.2 | Evaluable Analysis Set | 9 |
| | 4.2.3 | Use of analysis set | 9 |
| | 4.3 | Definition of Baseline | 9 |
| | 4.4 | Summary Statistics | 9 |
| | 4.5 | Significance Level | 10 |
| | 4.6 | Multiple Comparisons/Multiplicity | 10 |
| | 4.7 | Handling of Drop-outs, Missing Data and Outliers | 10 |
| | 4.8 | Adjustment for Covariates | 10 |
| | 4.9 | Multicentre Studies | 10 |
| | 4.10 | Examination of Subgroups | 10 |
| | 4.11 | Blind Review | |
| 5 | SU | BJECTS | 11 |
| | 5.1 | Subject Disposition | 11 |
| | 5.2 | Baseline Characteristics and Demographics | 11 |
| | 5.3 | Protocol Deviations | 11 |
| 6 | TR | EATMENT INFORMATION AND EXTENT OF EXPOSURE | 12 |
| | 6.1 | Active Treatment | 12 |
| | 6.2 | Prior and Concomitant Medications | 12 |




Study Code: BED-PSMA-101 CTC Project No: 213-22-2018

| 7 | STA | ATISTICAL METHODOLOGY | 13 |
|----|-------|---------------------------------------------------|----|
| | 7.1 | Primary Endpoint(s) Analysis | 13 |
| | 7.1.1 | Definition of endpoint(s) | 13 |
| | 7.2 | Main analytical approach | 14 |
| | 7.3 | Sensitivity analysis | 14 |
| | 7.4 | Supplementary analyses | 14 |
| | 7.5 | Presentation | 14 |
| | 7.6 | Secondary Endpoint(s) Analysis | 15 |
| | 7.6.1 | Definition of endpoint(s) | 15 |
| | 7.6.2 | Main analytical approach | 15 |
| | 7.6.3 | Sensitivity analysis | 15 |
| | 7.6.4 | Supplementary analyses | 15 |
| | 7.6.5 | Presentation | 15 |
| | 7.7 | Tertiary/Exploratory Endpoint(s) Analysis | 15 |
| | 7.8 | Discontinuation | 15 |
| | 7.9 | Other Analyses | 15 |
| | 7.10 | Interim Analysis | 15 |
| 8 | CH | ANGES FROM THE CSP | 16 |
| 9 | STA | ATISTICAL DELIVERABLES | 17 |
| 1( | 0 S | OFTWARE | 18 |
| 1 | 1 A | APPROVAL | 19 |
| 12 | 2 S | UPPORTIVE DOCUMENTATION | 20 |
| | 12.1 | Appendix 1 – List of Abbreviations | 20 |
| | 12.2 | Appendix 2 – Changes to Protocol-Planned Analyses | 22 |
| 1. | 3 S | TATISTICAL OUTPUTS LAYOUT | 23 |
| | 13.1 | Tables | 23 |
| | Sub | ect disposition | |
| | | nographic information | |
| | Pric | or and Concomitant Medications | 28 |
| | Stu | dy Drug Administration | 30 |
| | Preg | gnancy test | 31 |
| | | al Signs | |
| | ECO | G | 37 |
| | Safe | ety Laboratory – Clinical Chemistry | 51 |




Study Code: BED-PSMA-101 CTC Project No: 213-22-2018

| C Project No: 213-22-2018 | |
|---|---|
| Safety Laboratory – Coagulation | 63 |
| Safety Laboratory – Urine | 65 |
| Physical Examination | 70 |
| Gleason Grade and Score | 72 |
| Histopathology Results | 74 |
| Overview of Treatment Emergent Adverse Events | 75 |
| Overview of Pre-Treatment Adverse Events | 76 |
| Treatment Emergent Adverse Events by System Organ Class and Preferred Term | 77 |
| Pre-Treatment Adverse Events by System Organ Class and Preferred Term | 78 |
| 13.2 Listings | 79 |
| Discontinued Subjects | 79 |
| Protocol Deviations | 80 |
| Analysis Sets | 81 |
| Reason for Exclusion from Analysis Sets | 82 |
| Inclusion/Exclusion Exceptions | 83 |
| Demography | 84 |
| Virology Screen | 86 |
| Pregnancy Test | 87 |
| Medical History | 88 |
| Disease History and Therapies for PSA | 89 |
| PSA Laboratory Results (Historic Measurements) | 90 |
| Concomitant medications | 91 |
| Study Drug Administration | 92 |

Vital Signs9312-lead ECG Measurements94Safety Laboratory Results – Haematology95Safety Laboratory Results – Clinical Chemistry97Safety Laboratory Results – Urine100Physical Examinations101Gleason Grade and Score102Histopathology Results103Adverse Events104Serious Adverse Events105

Protocol Version No: 190222 BED CSP v1.0 final

Study Code: BED-PSMA-101 CTC Project No: 213-22-2018



5 (105)

### **VERSION HISTORY**

This Statistical Analysis Plan (SAP) for study BED-PSMA-101 is based on the protocol dated 22FEB2019.

**Table 1 SAP Version History Summary** 

| SAP version | Approval<br>Date | Changes | Rationale |
|-------------|------------------|---------|------------------|
| 1 | | NA | Original version |

### **INTRODUCTION**

This Statistical Analysis Plan (SAP) gives details regarding the statistical analyses and data presentation outlined in the final Clinical study protocol (CSP) for the study BED-PSMA-101. Any changes from the final CSP are given in Section 0.

BED-PSMA-101\_213-22-2018\_SAP\_v1.0\_30OCT2019


Study Code: BED-PSMA-101 CTC Project No: 213-22-2018



# 3 CLINICAL STUDY DETAILS

# 3.1 Clinical Study Objectives and Endpoints

| Objects | Estimands/Endpoints |
|---|---|
| Primary | |
| To assess the safety of a single<br>administration of <sup>18</sup> F-rhPSMA-7.3 in<br>healthy subjects and subjects with PCa. | Safety is the primary endpoint of the study and it will be assessed from data on the occurrence of one or more treatment-emergent AEs from the time of i.v. administration of <sup>18</sup> F-rhPSMA-7.3 throughout the study period, and changes in serum biochemistry, haematology, coagulation, urinalysis, vital signs, ECG, injection site status, and physical examination findings. |
| <ul> <li>To determine the biodistribution of <sup>18</sup>F following intravenous (i.v.) administration of <sup>18</sup>F-rhPSMA-7.3 and hence calculate the internal radiation dosimetry and the effective dose (ED) in healthy volunteers.</li> <li>To explore the optimization of PET imaging with <sup>18</sup>F-rhPSMA-7.3 injection in visualizing tumours in subjects with biopsy-proven PCa.</li> <li>To preform kinetic modelling on the distribution of <sup>18</sup>F-rhPSMA-7.3 in subjects with PCa.</li> <li>To use the kinetic modelling data to optimize protocol for future studies in subjects with PCa.</li> <li>To determine the <i>in vivo</i> Stability of <sup>18</sup>F-rhPSMA-7.3 injection by determining proportion of radioactive parent compound present over time.</li> </ul> | <ul> <li>Dosimetry estimates and cumulated radioactivity exposure by source region and the entire body including analysis of radioactivity in whole blood, plasma and excreted urine in healthy volunteers.</li> <li>Uptake of <sup>18</sup>Fr-h-PSMA-7.3 visualised by PET imaging compared to histopathology in subjects with PCa, if histopathology information is available.</li> <li>Use of kinetic modelling data to investigate distribution of <sup>18</sup>Frh-PSMA-7.3 in subjects with PCa.</li> <li>Use of kinetic modelling data to optimise the imaging protocol for future studies in subjects with PCA, by estimating <i>in vivo</i> <sup>18</sup>F radioactivity in PCa lesions</li> <li>Analysis of % of radioactive parent compound present in plasma over time in healthy volunteers and subjects with PCa. Relative proportions of radioactive tracer metabolites will be monitored, as well, if detected in significant amounts in the radio-HPLC analysis.</li> </ul> |
| Tertiary/Exploratory | |

BED-PSMA-101\_213-22-2018\_SAP\_v1.0\_30OCT2019


Study Code: BED-PSMA-101 CTC Project No: 213-22-2018



# 3.2 Clinical Study Design

This is a phase 1, open-label, single administration, healthy volunteer and patient study of a PET imaging agent performed at a single centre. The use of placebo, randomisation or blinding are not applicable in this study. Altogether 15 evaluable subjects are planned to participate in the trial: 6 healthy volunteer subjects (3 males and 3 females) and 9 patients with PCa (3 in each patient cohort). Additional subjects may be enrolled in order to end up with evaluable PET imaging data from 6 healthy volunteer subjects and 9 patients with PCa. Each subject will receive a single i.v. administration of <sup>18</sup>F-rhPSMA-7.3.

### 3.3 Statistical Hypotheses

No formal statistical hypotheses are stated. This study is exploratory in nature.

### 3.4 Number of Subjects

Fifteen (15) evaluable subjects will be included in the study: 6 healthy volunteer subjects (3 males, 3 females); 3 patients with high risk PCa, 3 patients with hormone sensitive metastatic PCa, and 3 patients with castration-resistant metastatic PCa. If an included subject's results are non-evaluable (see section 3.5 – Evaluability criteria), an additional subject may be included in the study to substitute for this.

#### 3.5 Evaluability criteria

Healthy Volunteer Evaluability Criteria:

The following criteria will be applied for evaluable healthy volunteers:

• Completion of scanning sessions I, II and III and collection of venous blood and urine analysis (as described in the Study Imaging Manual) to be able to undertake a calculation of the subject's internal radiation dosimetry.

Patient Evaluability Criteria:

The following criteria will be applied and if the patient is not evaluable for efficacy, an additional subject may be included in the study to substitute for the non-evaluable subject:

- Completion of scanning sessions I and II and collection of venous blood and urine analysis (as described in the Study Imaging Manual) to be able to perform kinetic modelling.
- At least one positive lesion on the <sup>18</sup>F-rhPSMA-7.3 scan.
- Cohort A only: Radical prostatectomy performed within 30 days of the <sup>18</sup>F-rhPSMA-7.3 scan. In case of a delay of the planned surgery by up to 2 days beyond this 30-day window, a subject may still be considered evaluable.


Study Code: BED-PSMA-101 CTC Project No: 213-22-2018



#### 3.6 Methods of Assigning Subject to IMP

The total duration of subject participation will be up to 52 days for each subject. The study consists of a screening period (up to 21 days), an IMP administration/PET imaging visit, a 24-hour post scan visit and a 30-day telephone contact. In case surgical prostatectomy is for some reason delayed in Cohort A patients scheduled for surgery, the participation of such subjects may be extended by up to two days to cover the surgery.

Subjects who sign the informed consent form (ICF) will enter the screening period of the study. A screening visit will take place within 21 days prior to the IMP administration/PET scan visit.

After the screening period, each subject will receive a single administration of IMP. The healthy volunteers will have 3 CT attenuation-correction scans, each followed by multiple whole-body (WB) PET acquisitions.

The subjects with PCa will have two CT attenuation-correction scans and dynamic PET imaging of the pelvic region (Cohort A) or the area with one or more metastases defined as representative target lesions (Cohorts B and C) for 45 min, followed by a 15 min break, and then multiple base of skull to mid-thigh PET acquisitions of up to 118 min p.i. The investigator will determine what the representative target lesions are in order to ensure that in the Cohort B and C patients all types of metastases, i.e. lymph node metastases, bone metastases, and soft tissue metastases, are represented on the dynamic images.

All subjects will attend a safety follow-up visit 24 hours (+/- 6 hours) after IMP administration and will be contacted by telephone 30 days (+/- 2 days; this may be extended further in Cohort A patients if the prostatectomy is delayed) after IMP administration to determine whether any AEs have occurred. Additional study visits will be arranged as needed for AE management. Any AEs will be followed up until resolution or stabilisation.

#### 3.7 Blinding

This is an open-label study; therefore, no blinding is needed in this study.


Study Code: BED-PSMA-101 CTC Project No: 213-22-2018



#### 4 STATISTICAL AND ANALYTICAL PLANS

#### 4.1 Sample Size Determination

Sufficient numbers of evaluable subjects have been planned to be included in the study in order to fulfil the study objectives, at the same time limiting the groups of healthy volunteer and patient volunteer subjects to the smallest informative numbers.

Altogether 15 evaluable subjects will be included in the study: 6 evaluable healthy volunteer subjects (3 males, 3 females), 3 evaluable subjects with high risk PCa (Cohort A), 3 evaluable subjects with hormone sensitive metastatic PCa (Cohort B), and 3 evaluable subjects with castration resistant metastatic disease (Cohort C).

### 4.2 Definition of Analysis Sets

### 4.2.1 Safety Analysis Set

The safety analysis set (SAF) will include all subjects who received any administration of the IMP.

### 4.2.2 Evaluable Analysis Set

Evaluable analysis set (EAS) will include all subjects who met all inclusion and exclusion criteria, received IMP, underwent PET/CT scans and met the scan evaluability criteria set.

### 4.2.3 Use of analysis set

The SAF will be used for safety evaluation. EAS will be used for the efficacy (i.e. secondary objectives) evaluations.

#### 4.3 Definition of Baseline

Baseline measurement is defined as the latest measurement prior to first dose of IMP at visit 2.

### 4.4 Summary Statistics

In general, all data collected will be presented with summary statistics and given in patient data listings. Summary statistics will include at least number of patients, mean, standard deviation, median, minimum and maximum for continuous data and frequency and percentage for categorical data. Table with summary statistics will be divided by treatment group, and assessment timepoint where applicable. Patient data listings will be sorted by treatment group, subject and timing of assessments.

The following treatment groups will be used for summary tables:

• Healthy Volunteers


Study Code: BED-PSMA-101 CTC Project No: 213-22-2018



- Patient Cohort A
- Patient Cohort B
- Patient Cohort C
- All Patient Cohorts (ie Cohorts A+B+C)
- All Cohorts (ie Healthy Volunteers + all patients)

### 4.5 Significance Level

Not applicable.

## 4.6 Multiple Comparisons/Multiplicity

No adjustment for multiple comparison/multiplicity will be performed, all significant statistical findings, must be reviewed for medical relevance.

## 4.7 Handling of Drop-outs, Missing Data and Outliers

Outliers will be included in summary tables and listings, and will not be handled separately in any analyses. No imputation of data will be performed.

### 4.8 Adjustment for Covariates

No adjustment for covariates will be performed.

#### 4.9 Multicentre Studies

No multicentre studies will be performed.

### 4.10Examination of Subgroups

No examination of subgroups will be performed.

#### 4.11Blind Review

Not applicable.


Study Code: BED-PSMA-101 CTC Project No: 213-22-2018



### 5 SUBJECTS

### **5.1 Subject Disposition**

The number of subjects that entered the study, withdrawn subjects, completed subjects and the number of subjects at each visit will be summarised by treatment.

# 5.2 Baseline Characteristics and Demographics

The following baseline characteristics will be summarised by treatment:

- Age
- Sex
- Ethnicity
- Race
- Use of nicotine
- Weight
- Height
- BMI

#### **5.3 Protocol Deviations**

A Protocol Deviation Log will be maintained for all protocol deviations, and the significance of each deviations will be assessed before database lock. All protocol deviations will be listed.

Protocol Version No: 190222 BED\_CSP\_v1.0\_final

Study Code: BED-PSMA-101 CTC Project No: 213-22-2018



### 6 TREATMENT INFORMATION AND EXTENT OF EXPOSURE

#### **6.1 Active Treatment**

The number of subjects who have been administered the IMP, the volume of undiluted IMP and the total administered activity will be summarised.

### 6.2 Prior and Concomitant Medications

Prior and concomitant medication data will be listed, and summarised by ATC name (Level 4 and Level 5, or the closest level). Prior and concomitant medications will be coded according to the World Health Organization (WHO) Anatomic Therapeutic Chemical (ATC) classification system.


Study Code: BED-PSMA-101 CTC Project No: 213-22-2018



#### 7 STATISTICAL METHODOLOGY

All parameters will be presented by treatment and assessment timepoint using summary statistics. Additional statistical analyses are specified below.

### 7.1 Primary Endpoint(s) Analysis

### 7.1.1 **Definition of endpoint(s)**

#### 7.1.1.1 Adverse events

All AEs will be summarised according to time of appearance (screening period and post-administration (=TEAE) AEs separately), following classification of the verbatim terms according to the Medical Dictionary for Regulatory Activities (MedDRA) dictionary. The number and percentage of subjects for all classified events will be presented according to System organ class (SOC) and Preferred term (PT) by subject group and overall.

Separate summaries will be presented for all AEs by subject and also for all AEs according to Seriousness, Severity and Relationship. For severity, if the subject has the same AE more than once but with different severities, the worst severity will be used for the summary. For relationship, if a subject has the same AE but if it is IMP-related at least once, then the AE will be considered as IMP-related in the summary.

If applicable, the following summaries by SOC and PT will also be produced.:

- Number of subjects with fatal AEs
- Number of subjects with AEs leading to study withdrawal
- The table will be sorted by alphabetic order.

The number and percentage of subjects with Injection site reaction during or within 4 h after IMP dosing will also be summarised, if applicable.

### 7.1.1.1 Vital signs

For blood pressure and pulse rate, descriptive statistics of actual values and of change from baseline will be used to summarise by treatment group and assessment timepoint. Baseline is defined as the value taken at visit 2, -5min to 0min, or this value is not available, then visit 2, -120min to -5min.

### 7.1.1.2 ECG resting 12-lead

ECG variables will be summarised according to actual values and change from baseline using summary statistics and will be presented by treatment group and assessment timepoint. Baseline is defined as the value taken at visit 2, -5 min to 0 min, or this value is not available, then visit 2, -120 min to -5 min.

### 7.1.1.3 Safety laboratory analyses

All haematology, clinical chemistry and coagulation laboratory tests will be summarised using descriptive statistics for actual values and change from baseline and presented by treatment group and assessment timepoint. Baseline is defined as the value taken at visit 2,


Study Code: BED-PSMA-101 CTC Project No: 213-22-2018



-5min to 0min, or this value is not available, then visit 2, -120min to -5min. All listings for safety laboratory will be sorted by laboratory parameter and then subject ID.

### 7.1.1.4 Physical examinations

Physical examination results will be categorically summarised as the number and percentage of subjects according to body system, treatment group and assessment timepoint.

#### 7.2 Main analytical approach

Summary statistics will include number of patients, mean, standard deviations, median, minimum and maximum for continuous data (mean and median will be presented to 1 additional decimal place relative to the collected data, and standard deviation will be presented to 2 additional decimal places related to the collected data) and frequency and percentage for categorical data.

### 7.3 Sensitivity analysis

No sensitivity analysis will be performed.

#### 7.4 Supplementary analyses

No supplementary analysis will be performed.

#### 7.5 Presentation

#### 7.5.1.1 Adverse Events

See tables and listings in Statistical Output Layout, section 13.

#### 7.5.1.2 Vital signs

See tables and listings in Statistical Output Layout, section 13.

#### 7.5.1.3 ECG resting 12-lead

See tables and listings in Statistical Output Layout, section 13.

#### 7.5.1.4 Safety laboratory analyses

See tables and listings in Statistical Output Layout, section 13.

#### 7.5.1.5 Physical examinations

See tables and listings in Statistical Output Layout, section 13.


Study Code: BED-PSMA-101 CTC Project No: 213-22-2018



### 7.6 Secondary Endpoint(s) Analysis

### 7.6.1 **Definition of endpoint(s)**

The biodistribution and dosimetry analyses in the Healthy Volunteers, and the kinetic modelling in the Patients, are described in the "BED-PSMA-101 Imaging Data Management Plan" written by Turku PET Centre. These analyses will be performed by Turku PET Centre in a separate report.

### 7.6.2 Main analytical approach

Not applicable.

# 7.6.3 Sensitivity analysis

No sensitivity analysis will be performed.

### 7.6.4 Supplementary analyses

No supplementary analysis will be performed.

#### 7.6.5 Presentation

Not applicable.

### 7.7 Tertiary/Exploratory Endpoint(s) Analysis

No tertiary/exploratory endpoints analysis will be performed.

#### 7.8 Discontinuation

Patients who discontinue from IMP treatment will be tabulated. The reason for discontinuation will be given. For discontinuation due to AE, the AEs will be given.

### 7.9 Other Analyses

No other analysis will be performed.

### 7.10Interim Analysis

No interim analysis will be performed.


Study Code: BED-PSMA-101 CTC Project No: 213-22-2018



### **CHANGES FROM THE CSP**

The following have been changed or added regarding to the CSP:

- FAS and PPS population have been taken away from the study. Decision from the sponsor, a protocol amendment will be written by sponsor.
- Categorically classified (Normal/Abnormal) results have been taken away from the sections 7.1.1.1 Vital signs and 7.1.1.2 ECG resting 12-lead. Decision from the sponsor.

BED-PSMA-101\_213-22-2018\_SAP\_v1.0\_30OCT2019


Study Code: BED-PSMA-101 CTC Project No: 213-22-2018



# 9 STATISTICAL DELIVERABLES

The following documents will be delivered:

- SAP
- Statistical analyses and summary tables


Study Code: BED-PSMA-101 CTC Project No: 213-22-2018



# 10 SOFTWARE

All statistical analyses will be performed using SAS Version 9.4 (SAS institute, Cary, NC).


Study Code: BED-PSMA-101 CTC Project No: 213-22-2018



# 11 APPROVAL

Issued by:

Fredrik Hansson, Director Biometrics

CTC Representative

11NOU2019

Date (dd-Mmm-yyyy)

Approved by:

Sponsor Representative

Date (dd-Mmm-yyyy)

05-NOV-2019


Study Code: BED-PSMA-101 CTC Project No: 213-22-2018



# 12 SUPPORTIVE DOCUMENTATION

# 12.1 Appendix 1 – List of Abbreviations

| Abbreviation of term | Explanation |
|----------------------|--------------------------------------------|
| ADL | Activities of daily living |
| ADR | Adverse drug reaction |
| AE | Adverse event |
| ATC | Anatomical-Therapeutic-Chemical |
| AUC | Area under the concentration by time curve |
| BMI | Body mass index |
| BP | Blood pressure |
| CA | Competent authority |
| CF | Clean File |
| $C_{\text{max}}$ | Maximum observed concentration |
| CRF | Case Report Form |
| CSP | Clinical study protocol |
| CT | Computed tomography |
| DM | Data management |
| EC | Ethics committee |
| ECG | Electrocardiography |
| ECOG | Eastern Cooperative Oncology Group |
| (e)CRF | (electronic) Case report form |
| ED | Effective dose |
| <sup>18</sup> F | Isotope of fluorine |
| FAS | Full Analysis Set |
| FSH | Follicle Stimulating Hormone |
| GCP | Good Clinical Practise |
| GDPR | General Data Protection Regulation |
| GLP | Good Laboratory Practise |
| GMP | Good Manufacturing Practise |
| HBsAg | Hepatitis B virus surface antigens |
| HCVAg | Hepatitis C virus antibodies |






Study Code: BED-PSMA-101 CTC Project No: 213-22-2018

HIVAgAb Human immunodeficiency virus antibodies

HR Heart rate

IC Informed consent

ICF Informed consent form
ISF Investigator's study file

IMP Investigational medicinal product

i.v. Intravenous

MBq Mega Becquerel

MCV Mean Corpuscular Volume

MCH Mean Corpuscular Haemoglobin

MedDRA Medical Dictionary for Regulatory Activities

mpMRI Multi-parametric MRI

mSv MilliSievert

OTC Over-the-counter
p.i. Post injection
PCa Prostate cancer

PET Positron Emission Tomography

PPS Per Protocol Set

PSA Prostate specific antigen

PSMA Prostate specific membrane antigen

PT Preferred term

RECIST Response Evaluation Criteria in Solid Tumours

SAE Serious adverse event
SAP Statistical Analysis Plan
SAS Statistical Analysis System

SAF Safety Analysis Set
SD Standard Deviation
SOC System Organ Class

SOP Standard operating procedure

SUSAR Suspected unexpected serious adverse reaction

SUV Standardized Uptake Value

SUVR Standardized Uptake Value Ratio


Study Code: BED-PSMA-101 CTC Project No: 213-22-2018



t½Elimination half-lifeTMFTrial Master FileTPCTurku PET CentreTRUSTransrectal ultrasound

# 12.2 Appendix 2 – Changes to Protocol-Planned Analyses


Study Code: BED-PSMA-101 CTC Project No: 213-22-2018



### 13 STATISTICAL OUTPUTS LAYOUT

# 13.1Tables

All tables will be grouped by: Healthy Volunteers, Cohort A, Cohort B, Cohort C, Cohort A+B+C and All Subjects.

Subject disposition

TABLE 14.1.1.1 SUBJECT DISPOSITION (ALL SUBJECTS)

| | Treatment A | Treatment B | Total |
|---------------------------------|-------------|-------------|-------|
| Screened subjects | XX | XX | XX |
| Subjects that entered the study | XX | xx | XX |
| Withdrawn subjects | XX | XX | XX |
| Completed subjects | XX | XX | XX |
| Included in SAF | XX | XX | XX |
| Included in EAS | XX | XX | XX |
| Subjects at Visit 1 (Screening) | XX | XX | XX |
| Subjects at Visit 2 | XX | XX | XX |
| Subjects at Visit 3 | XX | XX | XX |
| Subjects at Visit 4 | XX | xx | XX |


Study Code: BED-PSMA-101 CTC Project No: 213-22-2018



# Demographic information

#### TABLE 14.1.2.1 BASELINE CHARACTERISTICS AND DEMOGRAPHICS (EAS)

| | | Treatment A (N=xx) | Treatment B (N=xx) | Total (N=xx) |
|---|---|---|---|---|
| Age (years) | n | xx | XX | XX |
| | Mean (SD) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| | Median (Min, Max) | xx.x(x, xx) | xx.x(x, xx) | xx.x(x, xx) |
| Age Group (years) | <65 | xx(xx%) | xx(xx%) | xx(xx%) |
| | 65-<75 | xx(xx%) | xx(xx%) | xx(xx%) |
| | >=75 | xx(xx%) | xx(xx%) | xx(xx%) |
| Sex | Female | xx(xx%) | xx(xx%) | xx(xx%) |
| | Male | xx(xx%) | xx(xx%) | xx(xx%) |
| Ethnicity | Hispanic or Latino | xx(xx%) | xx(xx%) | xx(xx%) |
| | Non-Hispanic or Latino | xx(xx%) | xx(xx%) | xx(xx%) |
| | Not reported | xx(xx%) | xx(xx%) | xx(xx%) |
| Race | XXX | xx(xx%) | xx(xx%) | xx(xx%) |
| | XXX | xx(xx%) | xx(xx%) | xx(xx%)) |
| | XXX | xx(xx%) | xx(xx%) | xx(xx%) |
| | Not reported | xx(xx%) | xx(xx%) | xx(xx%) |
| Weight (kg) | n | xx | xx | XX |
| | Mean (SD) | xx.xx (x.xxx) | xx.xx (x.xxx) | xx.xx (x.xxx) |
| | Median (Min, Max) | xx.xx (x.x,.xx.x) | xx.xx(x.x,.xx.x) | xx.x(x.x,.xx.x) |
| Height (cm) | n | xx | XX | XX |
| | Mean (SD) | xx.x (x.x) | xx.x(x.x) | xx.x(x.x) |
| | Median (Min, Max) | xx.x(x, xx) | xx.x(x, xx) | xx.x(x, xx) |
| Body Mass Index (kg/m²) | n | xx | XX | XX |
| | Mean (SD) | xx.xx (x.xxx) | xx.xx (x.xxx) | xx.xx (x.xxx) |
| | Median (Min, Max) | xx.xx (x.xx, xx.x) | xx.x(x.xx, xx.x) | xx.x(x.xx, xx.x) |


CLINICAL TRIAL CONSULTANTS AB

Protocol Version No: 190222\_BED\_CSP\_v1.0\_final Study Code: BED-PSMA-101 CTC Project No: 213-22-2018

#### TABLE 14.1.2.2 BASELINE CHARACTERISTICS AND DEMOGRAPHICS (SAF)

| | | Treatment A (N=xx) | Treatment B (N=xx) | Total (N=xx) |
|---|---|---|---|---|
| Age (years) | n | xx | XX | XX |
| | Mean (SD) | xx.x (x.xx) | xx.x (x.xx) | xx.x(x.xx) |
| | Median (Min, Max) | xx.x(x, xx) | xx.x(x, xx) | xx.x(x, xx) |
| Age Group (years) | <65 | xx(xx%) | xx(xx%) | xx(xx%) |
| | 65-<75 | xx(xx%) | xx(xx%) | xx(xx%) |
| | >=75 | xx(xx%) | xx(xx%) | xx(xx%) |
| Sex | Female | Xx (xx.x%) | Xx (xx.x%) | Xx (xx.x%) |
| | Male | Xx (xx.x%) | Xx (xx.x%) | Xx (xx.x%) |
| Ethnicity | Hispanic or Latino | Xx (xx.x%) | Xx (xx.x%) | Xx (xx.x%) |
| | Non-Hispanic or Latino | Xx (xx.x%) | Xx (xx.x%) | Xx (xx.x%) |
| | Not reported | Xx (xx.x%) | Xx (xx.x%) | Xx (xx.x%) |
| Race | XXX | Xx (xx.x%) | Xx (xx.x%) | Xx (xx.x%) |
| | XXX | Xx (xx.x%) | Xx (xx.x%) | Xx (xx.x%) |
| | XXX | Xx (xx.x%) | Xx (xx.x%) | Xx (xx.x%) |
| | Not reported | Xx (xx.x%) | Xx (xx.x%) | Xx (xx.x%) |
| Weight (kg) | n | xx | XX | XX |
| | Mean (SD) | xx.xx (x.xxx) | xx.xx (x.xxx) | xx.xx (x.xxx) |
| | Median (Min, Max) | xx.xx (x.x,.xx.x) | xx.xx(x.x,.xx.x) | xx.x(x.x,.xx.x) |
| Height (cm) | N | xx | XX | XX |
| | Mean (SD) | xx.x (x.x) | xx.x(x.x) | xx.x(x.x) |
| | Median (Min, Max) | xx.x (x, xx) | xx.x(x, xx) | xx.x(x, xx) |
| Body Mass Index (kg/m²) | n | xx | XX | XX |
| | Mean (SD) | xx.xx (x.xxx) | xx.xx (x.xxx) | xx.xx (x.xxx) |
| | Median (Min, Max) | xx.xx (x.xx, xx.x) | xx.x(x.xx, xx.x) | xx.x(x.xx, xx.x) |
| ECOG | 0 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | 3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | 4 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

CONFIDENTIAL 25 (105) Protocol Version No: 190222\_BED\_CSP\_v1.0\_final

Study Code: BED-PSMA-101 CTC Project No: 213-22-2018

Medical/Surgical history

#### TABLE 14.1.3.1 MEDICAL HISTORY EVENTS BY SYSTEM ORGAN CLASS AND PREFERRED TERM (EAS)

| | Treatment A<br>N=xx | Treatment B<br>N=xx | Total<br>N=xx |
|---|---|---|---|
| System organ class<br>Preferred term | n(%) | n(%) | n(%) |
| Total | x(xx%) | x(xx%) | x(xx%) |
| Psychiatric disorders | x(xx%) | x(xx%) | x(xx%) |
| Anxiety | x(xx%) | x(xx%) | x(xx%) |
| Depression | x(xx%) | x(xx%) | x(xx%) |
| Insomnia | x(xx%) | x(xx%) | x(xx%) |
| Immune system disorders | x(xx%) | x(xx%) | x(xx%) |
| Hypersensitivity | x(xx%) | x(xx%) | x(xx%) |
| Seasonal allergy | x(xx%) | x(xx%) | x(xx%) |
| Metabolism and nutrition disorders | x(xx%) | x(xx%) | x(xx%) |
| Type 1 diabetes mellitus | x(xx%) | x(xx%) | x(xx%) |
| General disorders and administration site conditions | x(xx%) | x(xx%) | x(xx%) |
| Chronic fatigue syndrome | x(xx%) | x(xx%) | x(xx%) |
| Nervous system disorders | x(xx%) | x(xx%) | x(xx%) |
| Narcolepsy | x(xx%) | x(xx%) | x(xx%) |
| Reproductive system and breast disorders | x(xx%) | x(xx%) | x(xx%) |
| Premenstrual syndrome | x(xx%) | x(xx%) | x(xx%) |
| Respiratory, thoracic and mediastinal disorders | x(xx%) | x(xx%) | x(xx%) |
| Asthma | x(xx%) | x(xx%) | x(xx%) |
| Vascular disorders | x(xx%) | x(xx%) | x(xx%) |
| Hypertension | x(xx%) | x(xx%) | x(xx%) |

n, number of subjects;

Percentages are based on the number of subjects in the evaluable analysis set


CLINICAL TRIAL CONSULTANTS AB


Study Code: BED-PSMA-101 CTC Project No: 213-22-2018

#### TABLE 14.1.3.2 MEDICAL HISTORY EVENTS BY SYSTEM ORGAN CLASS AND PREFERRED TERM (SAF)

| | Treatment A N=xx | Treatment B<br>N=xx | Total<br>N=xx |
|---|---|---|---|
| System organ class<br>Preferred term | n(%) | n(%) | n(%) |
| Total | x(xx%) | x(xx%) | x(xx%) |
| Psychiatric disorders | x(xx%) | x(xx%) | x(xx%) |
| Anxiety | x(xx%) | x(xx%) | x(xx%) |
| Depression | x(xx%) | x(xx%) | x(xx%) |
| Insomnia | x(xx%) | x(xx%) | x(xx%) |
| Immune system disorders | x(xx%) | x(xx%) | x(xx%) |
| Hypersensitivity | x(xx%) | x(xx%) | x(xx%) |
| Seasonal allergy | x(xx%) | x(xx%) | x(xx%) |
| Metabolism and nutrition disorders | x(xx%) | x(xx%) | x(xx%) |
| Type 1 diabetes mellitus | x(xx%) | x(xx%) | x(xx%) |
| General disorders and administration site conditions | x(xx%) | x(xx%) | x(xx%) |
| Chronic fatigue syndrome | x(xx%) | x(xx%) | x(xx%) |
| Nervous system disorders | x(xx%) | x(xx%) | x(xx%) |
| Narcolepsy | x(xx%) | x(xx%) | x(xx%) |
| Reproductive system and breast disorders | x(xx%) | x(xx%) | x(xx%) |
| Premenstrual syndrome | x(xx%) | x(xx%) | x(xx%) |
| Respiratory, thoracic and mediastinal disorders | x(xx%) | x(xx%) | x(xx%) |
| Asthma | x(xx%) | x(xx%) | x(xx%) |
| Vascular disorders | x(xx%) | x(xx%) | x(xx%) |
| Hypertension | x(xx%) | x(xx%) | x(xx%) |

n, number of subjects;

Percentages are based on the number of subjects in the evaluable analysis set

BED-PSMA-101\_213-22-2018\_SAP\_v1.0\_30OCT2019





Study Code: BED-PSMA-101 CTC Project No: 213-22-2018

**Prior and Concomitant Medications** 

#### TABLE 14.1.4.1 PRIOR MEDICATION BY ATC LEVEL 4 AND 5 (SAF)

| | Treatment A<br>N=xx | | Total<br>N=xx |
|------------------|---------------------|--------|---------------|
| ATC Name Level 4 | | | |
| ATC Name Level 5 | n(%) | n(%) | n(%) |
| Total | x(xx%) | x(xx%) | x(xx%) |
| Level 4 | x(xx%) | x(xx%) | x(xx%) |
| Level 5 | x(xx%) | x(xx%) | x(xx%) |
| Level 5 | x(xx%) | x(xx%) | x(xx%) |
| Level 5 | x(xx%) | x(xx%) | x(xx%) |
| Level 4 | x(xx%) | x(xx%) | x(xx%) |
| Level 5 | x(xx%) | x(xx%) | x(xx%) |
| Level 5 | x(xx%) | x(xx%) | x(xx%) |

n, number of subjects;

Percentages are based on the number of subjects in the safety analysis set


CLINICAL TRIAL CONSULTANTS AB


Study Code: BED-PSMA-101 CTC Project No: 213-22-2018

#### TABLE 14.1.4.2 CONCOMITANT MEDICATION BY ATC LEVEL 4 AND 5 (SAF)

| | Treatment A<br>N=xx | Treatment B<br>N=xx | Total<br>N=xx |
|------------------|---------------------|---------------------|---------------|
| ATC Name Level 4 | | | |
| ATC Name Level 5 | n(%) | n(%) | n(%) |
| Total | x(xx%) | x(xx%) | x(xx%) |
| Level 4 | x(xx%) | x(xx%) | x(xx%) |
| Level 5 | x(xx%) | x(xx%) | x(xx%) |
| Level 5 | x(xx%) | x(xx%) | x(xx%) |
| Level 5 | x(xx%) | x(xx%) | x(xx%) |
| Level 4 | x(xx%) | x(xx%) | x(xx%) |
| Level 5 | x(xx%) | x(xx%) | x(xx%) |
| Level 5 | x(xx%) | x(xx%) | x(xx%) |

n, number of subjects;

Percentages are based on the number of subjects in the safety analysis set

BED-PSMA-101\_213-22-2018\_SAP\_v1.0\_30OCT2019

CLINICAL TRIAL CONSULTANTS AB


Study Code: BED-PSMA-101 CTC Project No: 213-22-2018

Study Drug Administration

#### TABLE 14.1.6 STUDY DRUG ADMINISTRATION (EAS)

| Description of<br>Planned Arm | | Visit<br>Name | N | Mean (SD) | Median<br>(Min, Max) | |
|---|---|---|---|---|---|---|
| Study Arm | <sup>18</sup> F-rhPSMA-7.3 | VISIT X | Х | x.xx (x.xx) | xx (x.x, x.x) | _ |





Study Code: BED-PSMA-101 CTC Project No: 213-22-2018

Pregnancy test

#### TABLE 14.1.6 PREGNANCY TEST RESULTS (EAS) – FEMALE SUBJECTS ONLY

| | | | Treatment A | Treatment B |
|--------------------|---------------|----------|-------------|-------------|
| Assessment | Visit<br>Name | Result | | |
| Post-Menopausal | Visit X | Yes | x(xx%)/x | x(xx%)/x |
| | | No | x(xx%)/x | x(xx%)/x |
| Surgically Sterile | Visit X | Yes | x(xx%)/x | x(xx%)/x |
| | | No | x(xx%)/x | x(xx%)/x |
| Pregnancy test | Visit X | Negative | x(xx%)/x | x(xx%)/x |
| | | Positive | x(xx%)/x | x(xx%)/x |

BED-PSMA-101\_213-22-2018\_SAP\_v1.0\_30OCT2019


CLINICAL TRIAL CONSULTANTS AB


Study Code: BED-PSMA-101 CTC Project No: 213-22-2018

Vital Signs

#### TABLE 14.2.1.1.1 VITAL SIGNS MEASUREMENTS, PULSE (SAF)

| | | | | | | TREATMENT<br>GROUP | Total |
|---|---|---|---|---|---|---|---|
| Assessment (unit) | Result Category | Visit Name | Planned Study Day of<br>Visit | Planned Time Point<br>Name | | | |
| Pulse Rate (beats/min) | Measured value | VISIT X | | | N | x | X |
| | | | | | Mean (SD) | xx.x (x.x) | xx.x(x.x) |
| | | | | | Median (Min, Max) | xx.x (xx, xx) | xx.x(xx, xx) |
| | Absolute change from baseline | VISIT X | | | N | x | x |
| baseine | | | | Mean (SD) | x.x (x.x) | x.x(x.x) | |
| | | | | | Median (Min, Max) | x.x(x, x) | x.x(x, x) |




#### TABLE 14.2.1.1.2 VITAL SIGNS MEASUREMENTS, BLOOD PRESSURE (SAF)

| Assessment (unit) | Result Category | Visit Name | Planned Study Day of<br>Visit | Planned Time Point<br>Name | | TREATMENT<br>GROUP | Total |
|---|---|---|---|---|---|---|---|
| Diastolic Blood | Measured value | VISIT X | VISIt | Name | N | | |
| Pressure (mmHg) | Measured value | VISI1 X | | | N<br>M (GD) | X | X |
| | | | | | Mean (SD) | xx.x (x.x) | xx.x (x.x) |
| | | | | | Median (Min, Max) | xx.x (xx, xx) | xx.x(xx, xx) |
| | | | | | | | ••• |
| Absolute chan baseline | Absolute change from | n VISIT X | | | N | X | X |
| | baseline | | | | Mean (SD) | x.x (x.x) | x.x(x.x) |
| | | | | | Median (Min, Max) | x.x(x, x) | x.x(x, x) |
| Systolic Blood Pressure | Measured value | VISIT X | | | N | X | x |
| (mmHg) | | | | | Mean (SD) | xxx.x (x.x) | xxx.x (x.x) |
| | | | | | Median (Min, Max) | xxx.x (xxx, xxx) | xxx.x (xxx, xxx) |
| | Absolute change from | VISIT X | | | N | x | x |
| | baseline | | | | Mean (SD) | x.x (x.x) | x.x (x.x) |
| | | | | | Median (Min, Max) | x.x(x, x) | x.x(x, x) |


CLINICAL TRIAL CONSULTANTS AB


#### TABLE 14.2.1.1.3 VITAL SIGNS MEASUREMENTS, BODY TEMPERATURE (SAF)

| | | | | | TREATMENT<br>GROUP | Total |
|---|---|---|---|---|---|---|
| Result Category | Visit Name | Planned Study Day of<br>Visit | Planned Time Point<br>Name | | | |
| Measured value | VISIT X | | | N | X | x |
| | | | | Mean (SD) | xx.xx (x.xx) | xx.x (x.x) |
| | | | | Median (Min, Max) | xx.xx (xx.x,<br>xx.x) | xx.x (xx, xx) |
| Absolute change from | VISIT X | | | N | x | X |
| baseline | | | | Mean (SD) | x.xx (x.xx) | x.xx (x.xx) |
| | | | | Median (Min, Max) | x.xx (x.x, x.x) | x.xx(x.x, x.x) |
| | Measured value | Measured value VISIT X Absolute change from VISIT X | Result Category Visit Name Visit Measured value VISIT X Absolute change from VISIT X | Result Category Visit Name Visit Name Measured value VISIT X Absolute change from VISIT X | Result Category Visit Name Visit Name Measured value VISIT X Mean (SD) Median (Min, Max) Absolute change from baseline VISIT X N Mean (SD) Median (Min, Max) | Result Category Visit Name Planned Study Day of Planned Time Point Visit Name N Measured value VISIT X N Median (SD) xx.xx (xx.x) Median (Min, Max) xx.xx (xx.x) Absolute change from baseline VISIT X Mean (SD) xx.xx (xx.x) Mean (SD) xx.xx (xx.x) xx.x) Mean (SD) xx.xx (xx.x) Mean (SD) xx.xx (xx.x) Mean (SD) xx.xx (xx.x) Mean (SD) xx.xx (xx.x) xx.xx (xx.x) Mean (SD) xx.xx (xx.x) xx.xx (xx.x) |


CLINICAL TRIAL CONSULTANTS AB


#### TABLE 14.2.1.1.4 VITAL SIGNS MEASUREMENTS, RESPIRATORY RATE (BREATHS/MIN) (SAF)

| | | | | | | TREATMENT<br>GROUP | Total |
|---|---|---|---|---|---|---|---|
| Assessment (unit) | Result Category | Visit Name | Planned Study Day of<br>Visit | Planned Time Point<br>Name | | | |
| Respiratory rate | Measured value | VISIT X | | | N | X | x |
| (breath/min) | | | | | Mean (SD) | xx.xx (x.xx) | xx.x (x.x) |
| | | | | | Median (Min, Max) | xx.xx (xx.x,<br>xx.x) | xx.x (xx, xx) |
| | Absolute change from | VISIT X | | | N | x | x |
| | baseline | | | | Mean (SD) | x.xx (x.xx) | x.xx (x.xx) |
| | | | | | Median (Min, Max) | x.xx (x.x, x.x) | x.xx(x.x, x.x) |




#### TABLE 14.2.1.2 VITAL SIGNS INTERPRETATIONS, (SAF)

| | | | | | TREATMENT<br>GROUP | Total |
|---|---|---|---|---|---|---|
| Assessment | Visit Name | Planned Study Day of<br>Visit | Planned Time Point<br>Name | Result | | |
| Pulse Rate (beats/min) | VISIT X | | | XXX | x(x%)/x | x(xx%)/x |
| | | | | ••• | | |
| Systolic Blood Pressure (mmHg) | VISIT X | | | xxx | x(x%)/x | x(xx%)/x |
| Diastolic Blood Pressure | VISIT X | | | XXX | x(x%)/x | x(xx%)/x |
| (mmHg) | | | | ••• | | |
| Temperature (C) | VISIT X | | | XXX | x(x%)/x | x(xx%)/x |
| Respiratory rate (breath/min) | VISIT X | | | xxx | x(x%)/x | x(xx%)/x |

CLINICAL TRIAL CONSULTANTS AB

Protocol Version No: 190222\_BED\_CSP\_v1.0\_final Study Code: BED-PSMA-101

CTC Project No: 213-22-2018

**ECG** 

#### TABLE 14.2.2.1.1 12-LEAD ECG MEASURMENTS, QRS DURATION (SAF)

| | | | | | | TREATMENT<br>GROUP | Total |
|---|---|---|---|---|---|---|---|
| Assessment (unit) | Result Category | Visit Name | Planned Study Day of<br>Visit | Planned Time Point<br>Name | | | |
| QRS Duration, | Measured value | VISIT X | | | N | X | X |
| Aggregate (ms) | | | | | Mean (SD) | xx.x (x.x) | xx.x(x.x) |
| | | | | | Median (Min, Max) | xx.x (xx, xx) | xx.x(xx, xx) |
| | Absolute change from baseline | VISIT X | | | N | x | x |
| | | | | | Mean (SD) | x.x (x.x) | x.x(x.x) |
| | | | | | Median (Min, Max) | x.x(x, x) | x.x(x, x) |


CTC Project No: 213-22-2018



#### TABLE 14.2.2.1.2 12-LEAD ECG MEASURMENTS, QT INTERVAL (SAF)

| | | | | | | TREATMENT<br>GROUP | Total |
|---|---|---|---|---|---|---|---|
| Assessment (unit) | Result Category | Visit Name | Planned Study Day of<br>Visit | Planned Time Point<br>Name | | | |
| QT Interval, Aggregate | Measured value | VISIT X | | | N | X | X |
| (ms) | | | | | Mean (SD) | xx.x (x.x) | xx.x(x.x) |
| | | | | | Median (Min, Max) | xx.x (xx, xx) | xx.x(xx, xx) |
| | Absolute change from baseline | VISIT X | | | N | x | x |
| | | | | | Mean (SD) | x.x (x.x) | x.x(x.x) |
| | | | | | Median (Min, Max) | x.x(x, x) | x.x(x, x) |


CLINICAL TRIAL CONSULTANTS AB


#### TABLE 14.2.2.1.3 12-LEAD ECG MEASURMENTS, QTCF INTERVAL (SAF)

| | | | | | | TREATMENT<br>GROUP | Total |
|---|---|---|---|---|---|---|---|
| Assessment (unit) | Result Category | Visit Name | Planned Study Day of<br>Visit | Planned Time Point<br>Name | | | |
| QTcF Interval, | Measured value | VISIT X | | | N | X | X |
| Aggregate (ms) | | | | | Mean (SD) | xx.x (x.x) | xx.x(x.x) |
| | | | | | Median (Min, Max) | xx.x (xx, xx) | xx.x(xx, xx) |
| | Absolute change from | VISIT X | | | N | x | x |
| | baseline | | | | Mean (SD) | x.x (x.x) | x.x (x.x) |
| | | | | | Median (Min, Max) | x.x (x, x) | x.x(x, x) |
| | | | | | ••• | | |


CLINICAL TRIAL CONSULTANTS AB


CTC Project No: 213-22-2018

### TABLE 14.2.2.1.4 12-LEAD ECG MEASURMENTS, PR INTERVAL (SAF)

| | | | | | | TREATMENT<br>GROUP | Total |
|---|---|---|---|---|---|---|---|
| Assessment (unit) | Result Category | Visit Name | Planned Study Day of<br>Visit | Planned Time Point<br>Name | | | |
| PR Interval, Aggregate | Measured value | VISIT X | | | N | X | X |
| (ms) | | | | | Mean (SD) | xx.x (x.x) | xx.x (x.x) |
| | | | | | Median (Min, Max) | xx.x (xx, xx) | xx.x (xx, xx) |
| | | | | | | | ••• |
| | Absolute change from | VISIT X | | | N | x | X |
| | baseline | | | | Mean (SD) | x.x (x.x) | x.x (x.x) |
| | | | | | Median (Min, Max) | x.x (x, x) | x.x(x, x) |
| | | | | | ••• | | ••• |


CLINICAL TRIAL CONSULTANTS AB


CTC Project No: 213-22-2018

#### TABLE 14.2.2.1.5 12-LEAD ECG MEASURMENTS, ECG MIN HEART RATE (SAF)

| | | | | | | TREATMENT<br>GROUP | Total |
|---|---|---|---|---|---|---|---|
| Assessment (unit) | Result Category | Visit Name | Planned Study Day of<br>Visit | Planned Time Point<br>Name | | | |
| ECG heart rate | Measured value | VISIT X | | | N | X | X |
| (beats/min) | | | | | Mean (SD) | xx.x (x.x) | xx.x(x.x) |
| | | | | | Median (Min, Max) | xx.x (xx, xx) | xx.x (xx, xx) |
| | Absolute change from | VISIT X | | | N | х | x |
| | baseline | | | | Mean (SD) | x.x (x.x) | x.x (x.x) |
| | | | | | Median (Min, Max) | x.x (x, x) | x.x(x, x) |
| | | | | | | | ••• |




#### TABLE 14.2.2.2 ECG INTERPRETATIONS (SAF)

| | | | | | TREATMENT<br>GROUP | Total |
|---|---|---|---|---|---|---|
| Assessment | Visit Name | Planned Study Day of<br>Visit | Planned Time Point<br>Name | Result | | |
| QRS Duration, Aggregate | VISIT X | | | XXX | x(x%)/x | x(xx%)/x |
| | | | | ••• | | |
| QT Interval, Aggregate | VISIT X | | | xxx | x(x%)/x | x(xx%)/x |
| | | | | ••• | | |
| QTcF Interval, Aggregate | VISIT X | | | xxx | x(x%)/x | x(xx%)/x |
| | | | | ••• | | |
| PR Interval, Aggregate | VISIT X | | | xxx | x(x%)/x | x(xx%)/x |
| | | | | ••• | | |
| ECG min heart rate (beats/min) | VISIT X | | | xxx | x(x%)/x | x(xx%)/x |


CLINICAL TRIAL CONSULTANTS AB


Study Code: BED-PSMA-101 CTC Project No: 213-22-2018

#### TABLE 14.2.3.1.1 SAFETY LABORATORY RESULTS, HAEMATOLOGY (SAF)

TREATMENT GROUP

| | | | | GROUP |
|---|---|---|---|---|
| Assessment (unit) | Result Category | Visit Name | | |
| Haemoglobin (g/L) | Measured value | VISIT X | N | x |
| | | | Mean (SD) | xxx.x (x.x) |
| | | | Median (Min, Max) | xxx.x (xxx, xxx) |
| | Absolute change from baseline | VISIT X | N | X |
| | | | Mean (SD) | x.x (x.x) |
| | | | Median (Min, Max) | x.x (xx, x) |

#### TABLE 14.2.3.1.2 SAFETY LABORATORY RESULTS, HAEMATOCRIT (SAF)

TREATMENT GROUP

| Result Category | Visit Name | | |
|---|---|---|---|
| Measured value | VISIT X | N | x |
| | | Mean (SD) | xxx.x (x.x) |
| | | Median (Min, Max) | xxx.x (xxx, xxx) |
| Absolute change from | VISIT X | N | x |
| baseline | | Mean (SD) | x.x (x.x) |
| | | Median (Min, Max) | x.x (xx, x) |
| | Measured value | Measured value VISIT X Absolute change from VISIT X | Measured value VISIT X Mean (SD) Median (Min, Max) Absolute change from baseline VISIT X N Mean (SD) Median (Min, Max) |

BED-PSMA-101\_213-22-2018\_SAP\_v1.0\_30OCT2019


**CLINICAL TRIAL CONSULTANTS AB** 


#### TABLE 14.2.3.1.3 SAFETY LABORATORY RESULTS, ERYTHROCYTES (SAF)

| TREAT | M | EN. | I. |
|-------|----|-----|----|
| GRO | MΠ | P | |

| | | | | GROUP |
|---|---|---|---|---|
| Assessment (unit) | Result Category | Visit Name | | |
| Erythrocytes (10^12/L) | Measured value | VISIT X | N | x |
| | | | Mean (SD) | xxx.x (x.x) |
| | | | Median (Min, Max) | xxx.x (xxx, xxx) |
| | Absolute change from | VISIT X | N | x |
| | baseline | | Mean (SD) | x.x (x.x) |
| | | | Median (Min, Max) | x.x (xx, x) |
| 7 | ГАВ <b>LE 14.2.3.1.4 SAFE</b> T | TY LABORATORY RE | SULTS, MCV (SAF) | |

#### TREATMENT GROUP

| Assessment (unit) | Result Category | Visit Name | | |
|---|---|---|---|---|
| MCV (/L) | Measured value | VISIT X | N | X |
| | | | Mean (SD) | xxx.x (x.x) |
| | | | Median (Min, Max) | xxx.x (xxx, xxx) |
| | Absolute change from baseline | VISIT X | N | x |
| | | | Mean (SD) | x.x (x.x) |
| | | | Median (Min, Max) | x.x (xx, x) |

BED-PSMA-101\_213-22-2018\_SAP\_v1.0\_30OCT2019


CLINICAL TRIAL CONSULTANTS AB


Study Code: BED-PSMA-101 CTC Project No: 213-22-2018

#### TABLE 14.2.3.1.5 SAFETY LABORATORY RESULTS, MCH (SAF)

| | | | | GROUP |
|---|---|---|---|---|
| Assessment (unit) | Result Category | Visit Name | | |
| MCH (pg) | Measured value | VISIT X | N | x |
| | | | Mean (SD) | xxx.x (x.x) |
| | | | Median (Min, Max) | xxx.x (xxx, xxx) |
| | Absolute change from | VISIT X | N | X |
| | baseline | | Mean (SD) | x.x (x.x) |
| | | | Median (Min, Max) | x.x (xx, x) |

#### TABLE 14.2.3.1.6 SAFETY LABORATORY RESULTS, PLATELETS (SAF)

TREATMENT GROUP

TREATMENT

| Assessment (unit) | Result Category | Visit Name | | |
|---|---|---|---|---|
| Platelets (10^9/L) | Measured value | VISIT X | N | X |
| | | | Mean (SD) | xxx.x (x.x) |
| | | | Median (Min, Max) | xxx.x (xxx, xxx) |
| | Absolute change from baseline | VISIT X | N | x |
| | | | Mean (SD) | x.x (x.x) |
| | | | Median (Min, Max) | x.x (xx, x) |


CLINICAL TRIAL CONSULTANTS AB


Study Code: BED-PSMA-101 CTC Project No: 213-22-2018

#### TABLE 14.2.3.1.7 SAFETY LABORATORY RESULTS, NEUTROPHILS (SAF)

TREATMENT GROUP

| | | | | 011001 |
|---|---|---|---|---|
| Assessment (unit) | Result Category | Visit Name | | |
| Neutrophils (10^9/L) | Measured value | VISIT X | N | x |
| | | | Mean (SD) | xxx.x (x.x) |
| | | | Median (Min, Max) | xxx.x (xxx, xxx) |
| | Absolute change from | VISIT X | N | X |
| baseline | | VISIT A | | A |
| | | | Mean (SD) | x.x(x.x) |
| | | | Median (Min, Max) | x.x (xx, x) |

#### TABLE 14.2.3.1.8 SAFETY LABORATORY RESULTS, EOSINOPHILS (SAF)

TREATMENT GROUP

| Assessment (unit) | Result Category | Visit Name | | |
|---|---|---|---|---|
| Eosinophils (10^9/L) | Measured value | VISIT X | N | x |
| | | | Mean (SD) | xxx.x (x.x) |
| | | | Median (Min, Max) | xxx.x (xxx, xxx) |
| | Absolute change from | VISIT X | N | x |
| | baseline | | Mean (SD) | x.x (x.x) |
| | | | Median (Min, Max) | x.x(xx, x) |


CLINICAL TRIAL CONSULTANTS AB


Study Code: BED-PSMA-101 CTC Project No: 213-22-2018

#### TABLE 14.2.3.1.9 SAFETY LABORATORY RESULTS, BASOPHILS (SAF)

| TREAT | M | EN. | I. |
|-------|----|-----|----|
| GRO | MΠ | P | |

| Assessment (unit) | Result Category | Visit Name | | |
|---|---|---|---|---|
| Basophils (10^9/L) | Measured value | VISIT X | N | x |
| | | | Mean (SD) | xxx.x (x.x) |
| | | | Median (Min, Max) | xxx.x (xxx, xxx) |
| | Absolute change from baseline | VISIT X | N | x |
| | | | Mean (SD) | x.x (x.x) |
| | | | Median (Min, Max) | x.x (xx, x) |

## TABLE 14.2.3.1.10 SAFETY LABORATORY RESULTS, LYMPHOCYTES (SAF)

## TREATMENT GROUP

| Assessment (unit) | Result Category | Visit Name | | |
|---|---|---|---|---|
| Lymphocytes (10^9/L) | Measured value | VISIT X | N | X |
| | | | Mean (SD) | xxx.x (x.x) |
| | | | Median (Min, Max) | xxx.x (xxx, xxx) |
| | Absolute change from baseline | VISIT X | N | x |
| | | | Mean (SD) | x.x (x.x) |
| | | | Median (Min, Max) | x.x (xx, x) |

BED-PSMA-101\_213-22-2018\_SAP\_v1.0\_30OCT2019


**CLINICAL TRIAL CONSULTANTS AB** 


CTC Project No: 213-22-2018

#### TABLE 14.2.3.1.12 SAFETY LABORATORY RESULTS, MONOCYTES (SAF)

TREATMENT GROUP

| | | | | GROOT |
|---|---|---|---|---|
| Assessment (unit) | Result Category | Visit Name | | |
| Monocytes (10^9/L) | Measured value | VISIT X | N | X |
| | | | Mean (SD) | xxx.x (x.x) |
| | | | Median (Min, Max) | xxx.x (xxx, xxx) |
| | Absolute change from baseline | VISIT X | N | x |
| | | | Mean (SD) | x.x (x.x) |
| | | | Median (Min, Max) | x.x (xx, x) |

BED-PSMA-101\_213-22-2018\_SAP\_v1.0\_30OCT2019


**CLINICAL TRIAL CONSULTANTS AB** 


CTC Project No: 213-22-2018

#### TABLE 14.2.3.1.2.1 SAFETY LABORATORY INTERPRETATIONS, HAEMATOLOGY (SAF)

| | | | | | TREATMENT<br>GROUP | Total |
|---|---|---|---|---|---|---|
| Assessment | Visit Name | Planned Study Day of<br>Visit | Planned Time<br>Point Name | Result | | |
| Haemoglobin | VISIT X | | | Normal/high/low | x(x%)/x | x(xx%)/x |
| | | | | | | ••• |
| Haematocrit | VISIT X | | | XXX | x(x%)/x | x(xx%)/x |
| | | | | | | ••• |
| Erythrocytes | VISIT X | | | XXX | x(x%)/x | x(xx%)/x |
| | | | | | | ••• |
| Leucocytes | VISIT X | | | xxx | x(x%)/x | x(xx%)/x |
| | | | | | | ••• |
| MCV | VISIT X | | | XXX | x(x%)/x | x(xx%)/x |
| | | | | | | ••• |
| MCH | VISIT X | | | xxx | x(x%)/x | x(xx%)/x |
| Platelets | VISIT X | | | xxx | x(x%)/x | x(xx%)/x |
| | | | | ••• | | ••• |


CLINICAL TRIAL CONSULTANTS AB


| x(x%)/x | x(xx%)/x |
|---------|-------------------------|
| | x(xx%)/x |
| x(x%)/x | x(xx%)/x |
| x(x%)/x | x(xx%)/x |
| x(x%)/x | x(xx%)/x |
| x(x%)/x | x(xx%)/x |
| | ••• |
| | x(x%)/x x(x%)/x x(x%)/x |

CONFIDENTIAL 50 (105) CLINICAL TRIAL CONSULTANTS AB


Study Code: BED-PSMA-101 CTC Project No: 213-22-2018

Safety Laboratory – Clinical Chemistry

#### TABLE 14.2.3.2.1 SAFETY LABORATORY RESULTS, ALKALINE (SAF)

## TREATMENT GROUP

| Assessment (unit) | Result Category | Visit Name | | |
|---|---|---|---|---|
| Alkaline Phosphatase | Measured value | VISIT X | N | X |
| (U/L) | | | Mean (SD) | xxx.x (x.x) |
| | | | Median (Min, Max) | xxx.x (xxx, xxx) |
| | Absolute change from baseline | VISIT X | N | x |
| | | | Mean (SD) | x.x (x.x) |
| | | | Median (Min, Max) | x.x (xx, x) |


CLINICAL TRIAL CONSULTANTS AB


Study Code: BED-PSMA-101 CTC Project No: 213-22-2018

#### TABLE 14.2.3.2.2 SAFETY LABORATORY RESULTS, ALANINE AMINOTRANSFERASE (SAF)

TREATMENT GROUP

| Assessment (unit) | Result Category | Visit Name | | |
|---|---|---|---|---|
| Alanine | Measured value | VISIT X | N | x |
| aminotransferase (U/L) | | | Mean (SD) | xxx.x (x.x) |
| | | | Median (Min, Max) | xxx.x (xxx, xxx) |
| | Absolute change from | VISIT X | N | x |
| | baseline | | Mean (SD) | x.x (x.x) |
| | | | Median (Min, Max) | x.x (xx, x) |

#### TABLE 14.2.3.2.3 SAFETY LABORATORY RESULTS, ASPARTATE AMINOTRANSFERASE (SAF)

TREATMENT GROUP

| Assessment (unit) | Result Category | Visit Name | | |
|---|---|---|---|---|
| Aspartate | Measured value | VISIT X | N | X |
| aminotransferase (U/L) | | | Mean (SD) | xxx.x (x.x) |
| | | | Median (Min, Max) | xxx.x (xxx, xxx) |
| | Absolute change from baseline | VISIT X | N | X |
| | | | Mean (SD) | x.x (x.x) |
| | | | Median (Min, Max) | x.x (xx, x) |
| | | | ••• | |


Study Code: BED-PSMA-101 CTC Project No: 213-22-2018

#### TABLE 14.2.3.2.4 SAFETY LABORATORY RESULTS, GAMMA-GLUTAMYL TRANSFERASE (SAF)

TREATMENT GROUP

| | | | | Olto 01 |
|---|---|---|---|---|
| Assessment (unit) | Result Category | Visit Name | | |
| Gamma-glutamyl | Measured value | VISIT X | N | x |
| transferase (U/L) | | | Mean (SD) | xxx.x (x.x) |
| | | | Median (Min, Max) | xxx.x (xxx, xxx) |
| | Absolute change from | VISIT X | N | x |
| | baseline | | Mean (SD) | x.x (x.x) |
| | | Median (Min, Max) | x.x (xx, x) | |

#### TABLE 14.2.3.2.5 SAFETY LABORATORY RESULTS, ALBUMIN (SAF)

TREATMENT GROUP

| Assessment (unit) | Result Category | Visit Name | | |
|---|---|---|---|---|
| Albumin (g/L) | Measured value | VISIT X | N | X |
| | | | Mean (SD) | xxx.x (x.x) |
| | | | Median (Min, Max) | xxx.x (xxx, xxx) |
| | Absolute change from | VISIT X | N | x |
| | baseline | | Mean (SD) x.x (x.x) | x.x (x.x) |
| | | | Median (Min, Max) | x.x (xx, x) |

BED-PSMA-101\_213-22-2018\_SAP\_v1.0\_30OCT2019


CLINICAL TRIAL CONSULTANTS AB


Study Code: BED-PSMA-101 CTC Project No: 213-22-2018

#### TABLE 14.2.3.2.6 SAFETY LABORATORY RESULTS, TOTAL PROTEIN (SAF)

| IK. | LA. | M | ΕN | 1 |
|-----|-----|-----|----|---|
| | GR | )II | P | |

| Assessment (unit) | Result Category | Visit Name | | |
|---|---|---|---|---|
| Total protein (g/L) | Measured value | VISIT X | N | x |
| | | | Mean (SD) | xxx.x (x.x) |
| | | | Median (Min, Max) | xxx.x (xxx, xxx) |
| | Absolute change from baseline | VISIT X | N | x |
| | | | Mean (SD) | x.x (x.x) |
| | | Median (Min, Max) | x.x (xx, x) | |

#### TABLE 14.2.3.2.7 SAFETY LABORATORY RESULTS, TOTAL BILIRUBIN (SAF)

## TREATMENT GROUP

| Assessment (unit) | Result Category | Visit Name | | |
|---|---|---|---|---|
| Total bilirubin (umol/L) | Measured value | VISIT X | N | X |
| | | | Mean (SD) | xxx.x (x.x) |
| | | | Median (Min, Max) | xxx.x (xxx, xxx) |
| | Absolute change from baseline | VISIT X | N x Mean (SD) x.x (x.x) | x |
| | | | | x.x (x.x) |
| | | | Median (Min, Max) | x.x (xx, x) |


CLINICAL TRIAL CONSULTANTS AB


Study Code: BED-PSMA-101 CTC Project No: 213-22-2018

#### TABLE 14.2.3.2.8 SAFETY LABORATORY RESULTS, CONJUGATED BILIRUBIN (SAF)

TREATMENT GROUP

| | | | | 011001 |
|---|---|---|---|---|
| Assessment (unit) | Result Category | Visit Name | | |
| Conjugated bilirubin | Measured value | VISIT X | N | x |
| (umol/L) | | | Mean (SD) | xxx.x (x.x) |
| | | | Median (Min, Max) | xxx.x (xxx, xxx) |
| | Absolute change from baseline | VISIT X | N | x |
| | baseine | Mean (SD) Median (Min, Max) | x.x (x.x) | |
| | | | Median (Min, Max) | x.x (xx, x) |

## TABLE 14.2.3.2.9 SAFETY LABORATORY RESULTS, CREATININE (SAF)

TREATMENT GROUP

| Assessment (unit) | Result Category | Visit Name | | |
|---|---|---|---|---|
| Creatinine (umol/L) | Measured value | VISIT X | N | X |
| | | | Mean (SD) | xxx.x (x.x) |
| | | | Median (Min, Max) | xxx.x (xxx, xxx) |
| | Absolute change from | VISIT X | N | x |
| | baseline | | Mean (SD) | x.x (x.x) |
| | | | Median (Min, Max) x.x | x.x (xx, x) |


CLINICAL TRIAL CONSULTANTS AB


Study Code: BED-PSMA-101 CTC Project No: 213-22-2018

#### TABLE 14.2.3.2.10 SAFETY LABORATORY RESULTS, UREA NITROGEN (BUN) (SAF)

TREATMENT GROUP

| | | | | GROOT |
|---|---|---|---|---|
| Assessment (unit) | Result Category | Visit Name | | |
| BUN (mmol/L) | Measured value | VISIT X | N | X |
| | | | Mean (SD) | xxx.x (x.x) |
| | | | Median (Min, Max) | xxx.x (xxx, xxx) |
| | | | ••• | |
| | Absolute change from baseline | VISIT X | N | x |
| | | Mean (SD)<br>Median (Min, Max | Mean (SD) | x.x (x.x) |
| | | | Median (Min, Max) | x.x (xx, x) |

#### TABLE 14.2.3.2.11 SAFETY LABORATORY RESULTS, CHLORIDE (SAF)

TREATMENT GROUP

| Assessment (unit) | Result Category | Visit Name | | |
|---|---|---|---|---|
| Chloride (mmol/L) | Measured value | VISIT X | N | x |
| | | | Mean (SD) | xxx.x (x.x) |
| | | | Median (Min, Max) | xxx.x (xxx, xxx) |
| | Absolute change from | VISIT X | N | x |
| baseline | | Mean (SD) | x.x (x.x) | |
| | | | Median (Min, Max) | x.x (xx, x) |


CLINICAL TRIAL CONSULTANTS AB


Study Code: BED-PSMA-101 CTC Project No: 213-22-2018

#### TABLE 14.2.3.2.12 SAFETY LABORATORY RESULTS, POTASSIUM (SAF)

| TREAT | M | EN. | I. |
|-------|----|-----|----|
| GRO | MΠ | P | |

| Assessment (unit) | Result Category | Visit Name | | |
|---|---|---|---|---|
| Potassium (mmol/L) | Measured value | VISIT X | N | x |
| | | | Mean (SD) | xxx.x (x.x) |
| | | | Median (Min, Max) | xxx.x (xxx, xxx) |
| | Absolute change from baseline | VISIT X | N | x |
| | | | Mean (SD) x.: | x.x (x.x) |
| | | Median (Min, Max) | x.x (xx, x) | |

## TABLE 14.2.3.2.13 SAFETY LABORATORY RESULTS, SODIUM (SAF)

## TREATMENT GROUP

| Assessment (unit) | Result Category | Visit Name | | |
|---|---|---|---|---|
| Sodium (mmol/L) | Measured value | VISIT X | N | X |
| | | | Mean (SD) | xxx.x (x.x) |
| | | | Median (Min, Max) | xxx.x (xxx, xxx) |
| | Absolute change from baseline | VISIT X N Mean (SD) | N | x |
| | | | x.x (x.x) | |
| | | | Median (Min, Max) | x.x (xx, x) |


CLINICAL TRIAL CONSULTANTS AB


Study Code: BED-PSMA-101 CTC Project No: 213-22-2018

#### TABLE 14.2.3.2.14 SAFETY LABORATORY RESULTS, C-REACTIVE PROTIEN (SAF)

TREATMENT GROUP

| | | | | 011001 |
|---|---|---|---|---|
| Assessment (unit) | Result Category | Visit Name | | |
| C-reactive protein | Measured value | VISIT X | N | x |
| (mg/L) | | | Mean (SD) | xxx.x (x.x) |
| | | | Median (Min, Max) | xxx.x (xxx, xxx) |
| | Absolute change from baseline | VISIT X | N | x |
| | | | Mean (SD) | x.x (x.x) |
| | | | Median (Min, Max) | x.x (xx, x) |
| | | | ••• | |

### TABLE 14.2.3.2.16 SAFETY LABORATORY RESULTS, FSH (FEMALE VOLUNTEERS ONLY) (SAF)

TREATMENT GROUP

| Assessment (unit) | Result Category | Visit Name | | |
|---|---|---|---|---|
| FSH (female volunteers | Measured value | VISIT X | N | X |
| only) (U/L) | | | Mean (SD) | xxx.x (x.x) |
| | | | Median (Min, Max) | xxx.x (xxx, xxx) |
| | Absolute change from baseline | VISIT X | N | x |
| | | | Mean (SD) | x.x (x.x) |
| | | | Median (Min, Max) | x.x (xx, x) |


CLINICAL TRIAL CONSULTANTS AB


BED-PSMA-101\_213-22-2018\_SAP\_v1.0\_30OCT2019

Study Code: BED-PSMA-101 CTC Project No: 213-22-2018

#### TABLE 14.2.3.2.17 SAFETY LABORATORY RESULTS, SERUM β-hCG-PREGNANCY TEST (FEMALE VOLUNTEERS ONLY) (SAF)

TREATMENT GROUP

| Assessment (unit) | Result Category | Visit Name | | |
|---|---|---|---|---|
| Serum β-hCG | Measured value | VISIT X | N | X |
| pregnancy test (female volunteers only) (U/L) | | | Mean (SD) | xxx.x (x.x) |
| | | | Median (Min, Max) | xxx.x (xxx, xxx) |
| | Absolute change from baseline | VISIT X | N | x |
| | | | Mean (SD) | x.x (x.x) |
| | | | Median (Min, Max) | x.x (xx, x) |


CLINICAL TRIAL CONSULTANTS AB


#### **TABLE 14.2.3.3.1 PSA (SAF)**

# TREATMENT GROUP

| | | | | GROUP |
|---|---|---|---|---|
| Assessment (unit) | Result Category | Visit Name | | |
| PSA (ng/mL)) | Measured value | VISIT X | N | x |
| | | | Mean (SD) | xxx.x (x.x) |
| | | | Median (Min, Max) | xxx.x (xxx, xxx) |
| | | | ••• | |
| | Absolute change from baseline | VISIT X | N | V |
| | | | IN | X |
| | | | Mean (SD) | x.x (x.x) |
| | | | Median (Min, Max) | x.x(xx, x) |


**CLINICAL TRIAL CONSULTANTS AB** 


CTC Project No: 213-22-2018

#### TABLE 14.2.3.2.2 SAFETY LABORATORY INTERPRETATIONS, CLINICAL CHEMISTRY (SAF)

| Assessment | Visit Name | Planned Study Day of<br>Visit | Planned Time Point<br>Name | Result | TREATMENT<br>GROUP | Total |
|---|---|---|---|---|---|---|
| Alkaline (ukat/L) | VISIT X | | | Low | x(x%)/x | x(x%)/x |
| ( ) | | | | Normal | x(x%)/x | x(x%)/x |
| | | | | High | x(x%)/x | x(x%)/x |
| Alanine aminotransferase (ukat/L) | VISIT X | | | XXX | x(x%)/x | x(xx%)/x |
| (uku/L) | | | | | | |
| Aspartate aminotransferase (ukat/L) | VISIT X | | | xxx | x(x%)/x | x(xx%)/x |
| ( | | | | | | |
| Gamma-glutamyl transferase<br>(ukat/L) | VISIT X | | | xxx | x(x%)/x | x(xx%)/x |
| (ukat/L) | | | | | | |
| Total bilirubin (unit) | VISIT X | | | xxx | x(x%)/x | x(xx%)/x |
| Conjugated bilirubin (unit) | VISIT X | | | xxx | x(x%)/x | x(xx%)/x |
| Creatinine (umol/L) | VISIT X | | | XXX | x(x%)/x | x(xx%)/x |


CLINICAL TRIAL CONSULTANTS AB


| | | | | | TREATMENT<br>GROUP | Total |
|---|---|---|---|---|---|---|
| Assessment | Visit Name | Planned Study Day of<br>Visit | Planned Time Point<br>Name | Result | | |
| | | | | ••• | | ••• |
| Urea nitrogen (BUN) (mmol/L) | VISIT X | | | xxx | x(x%)/x | x(xx%)/x |
| Potassium (mmol/L) | VISIT X | | | xxx | x(x%)/x | x(xx%)/x |
| Sodium (mmol/L) | VISIT X | | | XXX | x(x%)/x | x(xx%)/x |
| | | | | ••• | | ••• |
| C-reactive protein (mg/L) | VISIT X | | | XXX | x(x%)/x | x(xx%)/x |
| | | | | ••• | | ••• |
| FSH (female volunteers only) | VISIT X | | | XXX | x(x%)/x | x(xx%)/x |
| (U/L) | | | | | | |
| Serum β-hCG pregnancy test (female volunteers only) (U/L) | VISIT X | | | XXX | x(x%)/x | x(xx%)/x |
| (ternate volunteers only) (U/L) | | | | | | |


CLINICAL TRIAL CONSULTANTS AB


Study Code: BED-PSMA-101 CTC Project No: 213-22-2018

Safety Laboratory – Coagulation

#### TABLE 14.2.3.3.1 SAFETY LABORATORY RESULTS, COAGULATION (SAF)

| | | | | TREATMENT<br>GROUP |
|---|---|---|---|---|
| Assessment (unit) | Result Category | Visit Name | | |
| Activated Partial Thromboplastin Time | Measured value | VISIT X | N | x |
| (s) | | | Mean (SD) | xxx.x (x.x) |
| | | | Median (Min, Max) | xxx.x (xxx, xxx) |
| | Absolute change from baseline | VISIT X | N | X |
| | | | Mean (SD) | x.x (x.x) |
| | | | Median (Min, Max) | x.x(xx, x) |
| Prothrombin Intl. Normalized Ratio | Measured value | VISIT X | N | x |
| (ratio) | | | Mean (SD) | xxx.x (x.x) |
| | | | Median (Min, Max) | xxx.x (xxx, xxx) |
| | Absolute change from | VISIT X | N | x |
| | baseline | | Mean (SD) | x.x (x.x) |
| | | | Median (Min, Max) | x.x(xx, x) |


CLINICAL TRIAL CONSULTANTS AB


#### TABLE 14.2.3.3.2 SAFETY LABORATORY INTERPRETATIONS, COAGULATION (SAF)

| | | | | | TREATMENT<br>GROUP | Total |
|---|---|---|---|---|---|---|
| Assessment | Visit Name | Planned Study Day of<br>Visit | Planned Time Point<br>Name | Result | | |
| Activated Partial Thromboplastin Time | VISIT X | | | xxx<br> | x(x%)/x<br> | x(xx%)/x<br> |
| Prothrombin Intl. Normalized Ratio | VISIT X | | | xxx<br> | x(x%)/x<br> | x(xx%)/x<br> |

BED-PSMA-101\_213-22-2018\_SAP\_v1.0\_30OCT2019


**CLINICAL TRIAL CONSULTANTS AB** 


BED-PSMA-101\_213-22-2018\_SAP\_v1.0\_30OCT2019

Study Code: BED-PSMA-101 CTC Project No: 213-22-2018

Safety Laboratory – Urine

#### TABLE 14.2.3.4.1.1 SAFETY LABORATORY RESULTS, URINE - pH (SAF)

## TREATMENT

| | | | | | GROUP |
|---|---|---|---|---|---|
| | Assessment | Result Category | Visit Name | | |
| pН | | Measured value | VISIT X | N | x |
| | | | | Mean (SD) | xxx.x (x.x) |
| | | | | Median (Min, Max) | xxx.x (xxx, xxx) |
| | | Absolute change from | VISIT X | N | X |
| | | baseline | | Mean (SD) | x.x (x.x) |
| | | | | Median (Min, Max) | x.x (xx, x) |


CLINICAL TRIAL CONSULTANTS AB


Study Code: BED-PSMA-101 CTC Project No: 213-22-2018

#### TABLE 14.2.3.4.1.2 SAFETY LABORATORY RESULTS, URINE - RBC (SAF)

TREATMENT GROUP

| | | | | GROOT |
|---|---|---|---|---|
| Assessment | Result Category | Visit Name | | |
| RBC | Measured value | VISIT X | N | X |
| | | | Mean (SD) | xxx.x (x.x) |
| | | | Median (Min, Max) | xxx.x (xxx, xxx) |
| | Absolute change from baseline | VISIT X | N | x |
| | | | Mean (SD) | x.x (x.x) |
| | | | Median (Min, Max) | x.x (xx, x) |
| | | | | 1 |

#### TABLE 14.2.3.4.1.3 SAFETY LABORATORY RESULTS, URINE - WBC (SAF)

TREATMENT GROUP

| Assessment | Result Category | Visit Name | | |
|---|---|---|---|---|
| WBC | Measured value | VISIT X | N | x |
| | | | Mean (SD) | xxx.x (x.x) |
| | | | Median (Min, Max) | xxx.x (xxx, xxx) |
| | Absolute change from | VISIT X | N | x |
| | baseline | | Mean (SD) | x.x (x.x) |
| | | | Median (Min, Max) | x.x (xx, x) |


CLINICAL TRIAL CONSULTANTS AB


Study Code: BED-PSMA-101 CTC Project No: 213-22-2018

#### TABLE 14.2.3.4.1.4 SAFETY LABORATORY RESULTS, URINE - NITRITE (SAF)

TREATMENT GROUP

| Assessment | Result Category | Visit Name | | |
|---|---|---|---|---|
| Nitrite | Measured value | VISIT X | N | X |
| | | | Mean (SD) | xxx.x (x.x) |
| | | | Median (Min, Max) | xxx.x (xxx, xxx) |
| | Absolute change from baseline | VISIT X | N | x |
| | | | Mean (SD) | x.x (x.x) |
| | | | Median (Min, Max) | x.x (xx, x) |

#### TABLE 14.2.3.4.1.5 SAFETY LABORATORY RESULTS, URINE - PROTEIN (SAF)

TREATMENT GROUP

| Assessment | Result Category | Visit Name | | |
|---|---|---|---|---|
| Protein | Measured value | VISIT X | N | X |
| | | | Mean (SD) | xxx.x (x.x) |
| | | | Median (Min, Max) | xxx.x (xxx, xxx) |
| | Absolute change from | VISIT X | N | x |
| | baseline | | Mean (SD) | x.x (x.x) |
| | | | Median (Min, Max) | x.x (xx, x) |

BED-PSMA-101\_213-22-2018\_SAP\_v1.0\_30OCT2019


CLINICAL TRIAL CONSULTANTS AB


Study Code: BED-PSMA-101 CTC Project No: 213-22-2018

#### TABLE 14.2.3.4.1.6 SAFETY LABORATORY RESULTS, URINE - GLUCOSE (SAF)

TREATMENT GROUP

| Assessment | Result Category | Visit Name | | |
|---|---|---|---|---|
| Glucose | Measured value | VISIT X | N | X |
| | | | Mean (SD) | xxx.x (x.x) |
| | | | Median (Min, Max) | xxx.x (xxx, xxx) |
| | Absolute change from | VISIT X | N | x |
| | baseline | | Mean (SD) | x.x (x.x) |
| | | | Median (Min, Max) | x.x (xx, x) |

#### TABLE 14.2.3.4.1.7 SAFETY LABORATORY RESULTS, URINE KETONES (SAF)

TREATMENT GROUP

| Assessment | Result Category | Visit Name | | |
|---|---|---|---|---|
| Ketones | Measured value | VISIT X | N | X |
| | | | Mean (SD) | xxx.x (x.x) |
| | | | Median (Min, Max) | xxx.x (xxx, xxx) |
| | Absolute change from | VISIT X | N | x |
| | baseline | | Mean (SD) | x.x (x.x) |
| | | | Median (Min, Max) | x.x (xx, x) |

BED-PSMA-101\_213-22-2018\_SAP\_v1.0\_30OCT2019


CLINICAL TRIAL CONSULTANTS AB


#### TABLE 14.2.3.4.2 SAFETY LABORATORY INTERPRETATIONS, URINE (SAF)

| | | | | | TREATMENT<br>GROUP | Total |
|---|---|---|---|---|---|---|
| Assessment | Visit Name | Planned Study Day of<br>Visit | Planned Time Point<br>Name | Result | | |
| рН | VISIT X | | | XXX | x(x%)/x | x(xx%)/x |
| | | | | ••• | | ••• |
| RBC | VISIT X | | | xxx | x(x%)/x | x(xx%)/x |
| WBC | VISIT X | | | xxx | x(x%)/x | x(xx%)/x |
| | | | | ••• | | |
| Nitrite | VISIT X | | | xxx | x(x%)/x | x(xx%)/x |
| | | | | ••• | | ••• |
| Protein | VISIT X | | | xxx | x(x%)/x | x(xx%)/x |
| | | | | ••• | | ••• |
| Glucose | VISIT X | | | xxx | x(x%)/x | x(xx%)/x |
| Ketones | VISIT X | | | xxx | x(x%)/x | x(xx%)/x |
| | | | | ••• | | ••• |


Study Code: BED-PSMA-101 CTC Project No: 213-22-2018



Physical Examination

#### TABLE 14.2.4 PHYSICAL EXAMINATION (SAF)

| | | | TREATME<br>GROUP | NT<br>Total |
|--------------------------|---------|--------|------------------|-------------|
| Assessment | | | | |
| Head | Visit X | Normal | x(x%)/x | x(xx%)/x |
| Eyes, Ears, Nose, Throat | Visit X | Normal | x(x%)/x | x(xx%)/x |
| | | | | ••• |
| Cardiovascular | Visit X | Normal | x(x%)/x | x(xx%)/x |
| Respiratory | Visit X | Normal | x(x%)/x | x(xx%)/x |
| Musculoskeletal | Visit X | Normal | x(x%)/x | x(xx%)/x |
| Gastrointestinal | Visit X | Normal | x(x%)/x | x(xx%)/x |
| Hepatic | Visit X | Normal | x(x%)/x | x(xx%)/x |


CLINICAL TRIAL CONSULTANTS AB


| | | | TREATMENT GROUP | Total |
|--------------|---------|--------|-----------------|----------|
| Assessment | | | | |
| Psyche | Visit X | Normal | x(x%)/x | x(xx%)/x |
| | | | | ••• |
| Endocrine | Visit X | Normal | x(x%)/x | x(xx%)/x |
| | | | ••• | ••• |
| Dermatologic | Visit X | Normal | x(x%)/x | x(xx%)/x |
| Lymph nodes | Visit X | Normal | x(x%)/x | x(xx%)/x |





Study Code: BED-PSMA-101 CTC Project No: 213-22-2018

Gleason Grade and Score

#### TABLE 14.2.9 GLEASON GRADE AND SCORE, (PATIENT ONLY)

| | | | Patient only |
|-----------------|---------|-------|--------------|
| Assessment | Visit | Grade | |
| Primary Grade | Visit X | 1 | x(x%)/x |
| | | 2 | x(x%)/x |
| | | 3 | x(x%)/x |
| | | 4 | x(x%)/x |
| | | 5 | x(x%)/x |
| Secondary Grade | Visit X | 1 | x(x%)/x |
| | | 2 | x(x%)/x |
| | | 3 | x(x%)/x |
| | | 4 | x(x%)/x |
| | | 5 | x(x%)/x |
| | | ••• | ••• |
| Tertiary Grade | Visit X | 1 | x(x%)/x |
| | | 2 | x(x%)/x |
| | | 3 | x(x%)/x |
| | | 4 | x(x%)/x |
| | | 5 | x(x%)/x |
| | | | ••• |
| Gleason Grade | Visit X | 1 | x(x%)/x |
| | | 2 | x(x%)/x |

CLINICAL TRIAL CONSULTANTS AB


| | | | Patient only |
|------------|-------|-----|--------------|
| Assessment | Visit | Gra | de |
| | • | 3 | x(x%)/x |
| | | 4 | x(x%)/x |
| | | 5 | x(x%)/x |
| | | | x(x%)/x |





Study Code: BED-PSMA-101 CTC Project No: 213-22-2018

Histopathology Results

TABLE 14.2.10 HISTOPATHOLOGY RESULTS, (PATIENT ONLY)

BED-PSMA-101\_213-22-2018\_SAP\_v1.0\_30OCT2019


Study Code: BED-PSMA-101 CTC Project No: 213-22-2018



# Overview of Treatment Emergent Adverse Events

#### TABLE 14.3.1.1.1 OVERVIEW OF TREATMENT EMERGENT ADVERSE EVENTS, EAS

| | Treatment A<br>N=XX | Treatment B<br>N=XX | Total<br>N=XX |
|---|---|---|---|
| | n(%) | n(%) | n(%) |
| Any TEAE | x(xx%) | x(xx%) | x(xx%) |
| Any IMP-related TEAE | x(xx%) | x(xx%) | x(xx%) |
| Any SAE | x(xx%) | x(xx%) | x(xx%) |
| Any IMP-related SAE | x(xx%) | x(xx%) | x(xx%) |
| Any AE leading to withdrawal | x(xx%) | x(xx%) | x(xx%) |
| Any AE leading to death | x(xx%) | x(xx%) | x(xx%) |
| Severity | | | |
| Mild | x(xx%) | x(xx%) | x(xx%) |
| Moderate | x(xx%) | x(xx%) | x(xx%) |
| Sever | x(xx%) | x(xx%) | x(xx%) |

n, number of subjects; m, number of events

Percentages are based on the number of subjects in the treatment period included in the evaluable analysis set.

Adverse events that occurred during follow-up are omitted from summary.

BED-PSMA-101 213-22-2018 SAP v1.0 30OCT2019





Study Code: BED-PSMA-101 CTC Project No: 213-22-2018

Overview of Pre-Treatment Adverse Events

#### TABLE 14.3.1.1.2 OVERVIEW OF PRE-TREATMENT ADVERSE EVENTS, SAF

| | Treatment A N=XX | Treatment B<br>N=XX | Total<br>N=XX |
|---|---|---|---|
| | n(%) | n(%) | n(%) |
| Any TEAE | x(xx%) | x(xx%) | x(xx%) |
| Any IMP-related TEAE | x(xx%) | x(xx%) | x(xx%) |
| Any SAE | x(xx%) | x(xx%) | x(xx%) |
| Any IMP-related SAE | x(xx%) | x(xx%) | x(xx%) |
| Any AE leading to withdrawal | x(xx%) | x(xx%) | x(xx%) |
| Any AE leading to death | x(xx%) | x(xx%) | x(xx%) |
| Severity | | | |
| Mild | x(xx%) | x(xx%) | x(xx%) |
| Moderate | x(xx%) | x(xx%) | x(xx%) |
| Sever | x(xx%) | x(xx%) | x(xx%) |
| Relationship | | | |
| Not related | x(xx%) | x(xx%) | x(xx%) |
| Related | x(xx%) | x(xx%) | x(xx%) |
| Not applicable | x(xx%) | x(xx%) | x(xx%) |

n, number of subjects;

Percentages are based on the number of subjects in the treatment period included in the evaluable analysis set.

Adverse events that occurred during follow-up are omitted from summary.

BED-PSMA-101\_213-22-2018\_SAP\_v1.0\_30OCT2019





Study Code: BED-PSMA-101 CTC Project No: 213-22-2018

Treatment Emergent Adverse Events by System Organ Class and Preferred Term

#### TABLE 14.3.1.2.1 TREATMENT EMERGENT ADVERSE EVENTS BY SYSTEM ORGAN CLASS AND PREFERRED TERM, EAS

| | Treatment A<br>N=XX | Treatment B<br>N=XX | Total<br>N=XX |
|---|---|---|---|
| System organ class<br>Preferred term | n(%) | n(%) | n(%) |
| Gastrointestinal disorders | x(xx%) | x(xx%) | x(xx%) |
| Dry mouth | x(xx%) | x(xx%) | x(xx%) |
| Gingival blister | x(xx%) | x(xx%) | x(xx%) |
| Lip pain | x(xx%) | x(xx%) | x(xx%) |
| Nausea | x(xx%) | x(xx%) | x(xx%) |
| Infections and infestations | x(xx%) | x(xx%) | x(xx%) |
| Diarrhoea infectious | x(xx%) | x(xx%) | x(xx%) |
| Gastroenteritis viral | x(xx%) | x(xx%) | x(xx%) |
| Influenza | x(xx%) | x(xx%) | x(xx%) |
| Nasopharyngitis | x(xx%) | x(xx%) | x(xx%) |
| Nervous system disorders | x(xx%) | x(xx%) | x(xx%) |
| Dizziness | x(xx%) | x(xx%) | x(xx%) |

n, number of subjects;

Percentages are based on the number of subjects in the treatment period included in the evaluable analysis set.

Adverse events that occurred during follow-up are omitted from summary.

BED-PSMA-101 213-22-2018 SAP v1.0 30OCT2019


Study Code: BED-PSMA-101 CTC Project No: 213-22-2018



Pre-Treatment Adverse Events by System Organ Class and Preferred Term

#### TABLE 14.3.1.2.2 PRE-TREATMENT ADVERSE EVENTS BY SYSTEM ORGAN CLASS AND PREFERRED TERM, EAS

| | Treatment A<br>N=XX | Treatment B<br>N=XX | Total<br>N=XX |
|---|---|---|---|
| System organ class<br>Preferred term | n(%) | n(%) | n(%) |
| Gastrointestinal disorders | x(xx%) | x(xx%) | x(xx%) |
| Dry mouth | x(xx%) | x(xx%) | x(xx%) |
| Gingival blister | x(xx%) | x(xx%) | x(xx%) |
| Lip pain | x(xx%) | x(xx%) | x(xx%) |
| Nausea | x(xx%) | x(xx%) | x(xx%) |
| Infections and infestations | x(xx%) | x(xx%) | x(xx%) |
| Diarrhoea infectious | x(xx%) | x(xx%) | x(xx%) |
| Gastroenteritis viral | x(xx%) | x(xx%) | x(xx%) |
| Influenza | x(xx%) | x(xx%) | x(xx%) |
| Nasopharyngitis | x(xx%) | x(xx%) | x(xx%) |
| Nervous system disorders | x(xx%) | x(xx%) | x(xx%) |
| Dizziness | x(xx%) | x(xx%) | x(xx%) |

n, number of subjects;

Percentages are based on the number of subjects in the treatment period included in the evaluable analysis set.

Adverse events that occurred during follow-up are omitted from summary.

BED-PSMA-101\_213-22-2018\_SAP\_v1.0\_30OCT2019


Study Code: BED-PSMA-101 CTC Project No: 213-22-2018



# 13.2Listings

**Discontinued Subjects** 

### LISTING 16.2.1.1 DISCONTINUED SUBJECTS (ALL SUBJECTS)

| Description of<br>Planned Arm | Unique Subject<br>Identifier | Date of<br>discontinuation<br>(Study Day) | Reason for discontinuation | Standardised term for reason for discontinuation |
|---|---|---|---|---|
| Study Arm | Subject ID | YYYY-MM-DD<br>(XX) | Disposition Event | Disposition Event |

BED-PSMA-101\_213-22-2018\_SAP\_v1.0\_30OCT2019

**CLINICAL TRIAL CONSULTANTS AB** 


CTC Project No: 213-22-2018

# Protocol Deviations

### LISTING 16.2.2. PROTOCOL DEVIATIONS (ALL SUBJECTS)

| Description of Planned<br>Arm | Subject Identifier for the Study | Sequence Number | Protocol Deviation Term | | Other Action Taken |
|---|---|---|---|---|---|
| Study Arm | Subject ID | х | Deviation Term | Action Term | |


Study Code: BED-PSMA-101 CTC Project No: 213-22-2018

Analysis Sets



### LISTING 16.2.3.1 ANALYSIS SETS (ALL SUBJECTS)

| Description of<br>Planned Arm | Subject<br>Identifier for<br>the Study | Evaluable<br>Analysis Set | Safety<br>Analysis<br>Set |
|---|---|---|---|
| Study Arm | Subject ID | Y/N | Y/N |
| | ••• | | |

BED-PSMA-101\_213-22-2018\_SAP\_v1.0\_30OCT2019




Study Code: BED-PSMA-101 CTC Project No: 213-22-2018



Reason for Exclusion from Analysis Sets

BED-PSMA-101\_213-22-2018\_SAP\_v1.0\_30OCT2019

### LISTING 16.2.3.2 REASON FOR EXCLUSION FROM ANALYSIS SETS (ALL SUBJECTS)

| Description of<br>Planned Arm | Subject Identifier for the Study | Population | Reason for Exclusion |
|---|---|---|---|
| Study Arm | Subject ID | EAS/SAF | Reason |
| | | | ••• |


**CLINICAL TRIAL CONSULTANTS AB** 


CTC Project No: 213-22-2018

Inclusion/Exclusion Exceptions

### LISTING 16.2.3.3 INCLUSION/EXCLUSION EXPECTIONS (ALL SUBJECTS)

| Description of<br>Planned Arm | Subject<br>Identifier for<br>the Study | Date/Time of<br>Collection (Study<br>Day) | Inclusion/Exclusion<br>Category | Inclusion/Exclusion Criterion | I/E Criterion<br>Result in Std<br>Format |
|---|---|---|---|---|---|
| Study Arm | Subject ID | YYYY-MM-DD (xx) | Exclusion | Exclusion Criterion | Y/N |

BED-PSMA-101\_213-22-2018\_SAP\_v1.0\_30OCT2019

CLINICAL TRIAL CONSULTANTS AB


CTC Project No: 213-22-2018

Demography

### LISTING 16.2.4.1. DEMOGRAPHIC DATA (SAF)

| Description<br>of Planned<br>Arm | Subject<br>Identifier for<br>the Study | Age | Sex | Ethnicity | Race | Use of Nicotine |
|---|---|---|---|---|---|---|
| Study Arm | Subject ID | XX | M/F | xxx | XXX | Y/N |

BED-PSMA-101\_213-22-2018\_SAP\_v1.0\_30OCT2019


Study Code: BED-PSMA-101 CTC Project No: 213-22-2018



Alcohol and Drug Abuse During Study Period

BED-PSMA-101\_213-22-2018\_SAP\_v1.0\_30OCT2019

### LISTING 16.2.4.3 ALCOHOL AND DRUG ABUSE DURING STUDY (SAF)

| Description of Planned Arm | Subject<br>Identifier for the<br>Study | e Visit<br>Name | Date/Time of Alcohol Test<br>(Study Day) | Alcohol Test Result | Date/Time of Drug Test<br>(Study Day) | Drug Test Result |
|---|---|---|---|---|---|---|
| Study Arm | Subject ID | Visit x | YYYY-MM-DD (XX) | Negative/Positive | YYYY-MM-DD (XX) | Negative/Positive |
| Study Arm | Subject ID | Visit x | YYYY-MM-DD (XX) | Negative/Positive | YYYY-MM-DD (XX) | Negative/Positive |




CTC Project No: 213-22-2018

Virology Screen

### LISTING 16.2.4.4 VIROLOGY SCREEN, ECOG (SAF)

| Description of<br>Planned Arm | Subject<br>Identifier for the<br>Study | Visit Name | Date/Time of<br>Virology Screen<br>(Study Day) | Test Result |
|---|---|---|---|---|
| Study Arm | Subject ID | Visit 1 | YYYY-MM-DD (xx) | Negative/Positive |

BED-PSMA-101\_213-22-2018\_SAP\_v1.0\_30OCT2019




CTC Project No: 213-22-2018

Pregnancy Test

### LISTING 16.2.4.5 PREGNANCY TEST RESULTS (SAF) – FEMALE SUBJECTS ONLY

| Description of<br>Planned Arm | Subject<br>Identifier for the<br>Study | Visit Name | Post-menopausa | l Surgically<br>Sterile | Lab Test or<br>Examination<br>Name | Date/Time of<br>Pregnancy Test<br>(Study Day) | Type of Pregnancy<br>Test | Test Result |
|---|---|---|---|---|---|---|---|---|
| Study Arm | Subject ID | Visit 1 | Yes/No | Yes/No | Pregnancy test | YYYY-MM-DD (xx) | Urine / Serum | Negative/Positive |


**CLINICAL TRIAL CONSULTANTS AB** 


CTC Project No: 213-22-2018

Medical History

### LISTING 16.2.5.1 MEDICAL HISTORY (SAF)

| Description of<br>Planned Arm | Subject<br>Identifier for<br>the Study | Reported Term for the Medical History | Dictionary-Derived<br>Term | Body System or Organ<br>Class | Start Date of Medical<br>History Event (Study<br>Day) | End Date of Medical<br>History Event (Study<br>Day) |
|---|---|---|---|---|---|---|
| Study Arm | Subject ID | Medical Term | Term | System | YYYY-MM-DD (XX) | YYYY-MM-DD (XX) |


CLINICAL TRIAL CONSULTANTS AB


Study Code: BED-PSMA-101 CTC Project No: 213-22-2018

Disease History and Therapies for PSA

#### LISTING 16.2.5.2. PROSTATE CANCER HISTORY

| Description of Planned Arm | Subject Identifier for the Study | Date of initial<br>prostate cancer<br>diagnosis<br>(Study Day) | Therapy | Therapy<br>Name | Dose | Unit | Route | Start Date<br>(Study Day) | End Date<br>(Study Day) | Ongoing |
|---|---|---|---|---|---|---|---|---|---|---|
| Study Arm | Subject ID | YYYY-MM-<br>DD (XX) | XX | xx | XX | xx | XX | XX | XX | XX |
| ••• | ••• | | | | | | | | | |

### LISTING 16.2.5.3. DISEASE THERAPIES FOR PSA (ONLY PATIENT POPULAITON)

| Description of Planned Arm | Subject Identifier for the Study | Sequence<br>Number | Start Date/Time of<br>Medical History Event | End Date/Time of<br>Medical History Event | Study Day of Start<br>of Observation | Study Day of End of Observation | PSA value | PSA baseline |
|---|---|---|---|---|---|---|---|---|
| Study Arm | Subject ID | X | YYYY-MM-DD | YYYY-MM-DD | xxx | XXX | х | Y/N |
| | ••• | | ••• | ••• | ••• | ••• | | |

BED-PSMA-101\_213-22-2018\_SAP\_v1.0\_30OCT2019


**CLINICAL TRIAL CONSULTANTS AB** 


Study Code: BED-PSMA-101 CTC Project No: 213-22-2018

PSA Laboratory Results (Historic Measurements)

### LISTING 16.2.5.3. PSA LABORATORY RESULTS (HISTORIC MEASUREMENTS) (ONLY PATIENT POPULAITON)

| Description of<br>Planned Arm | Subject<br>Identifier for the<br>Study | Date<br>of PSA (Study Day) | Result (ng/mL) |
|---|---|---|---|
| Study Arm | Subject ID | YYYY-MM-DD<br>(XX) | XX.X |


BED-PSMA-101\_213-22-2018\_SAP\_v1.0\_30OCT2019

**CLINICAL TRIAL CONSULTANTS AB** 


CTC Project No: 213-22-2018

Concomitant medications

### LISTING 16.2.6.1 CONCOMITANT MEDICATIONS, INDICATIONS (SAF)

#### TREATMENT GROUP = XXX

| Subject<br>Identifier for<br>the Study | Reported<br>Name of<br>Drug, Med,<br>or Therapy | Standardized<br>Medication Name<br>ATC Level 5 (ATC<br>Level 4) | Medication Class<br>Code | Category for<br>Medication | Details | Dose<br>Description | Dose<br>Units | Route of Administration | Dosing<br>Frequency<br>per Interval | Dose<br>Form | Start Date (Study<br>Day) | End Date (Study Day) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject ID | Xxx | xxx (xxx) | XX | Medical/ surgical history | MH/AE term | xx | mg | Oral | Daily | Tablet | YYYY-MM-DD<br>(XX) | YYYY-MM-DD<br>(XX) |
| ••• | | | | | | | | | | | | |


CLINICAL TRIAL CONSULTANTS AB


Study Code: BED-PSMA-101 CTC Project No: 213-22-2018

# Study Drug Administration

### LISTING 16.2.7. ADMINISTRATION OF (SAF) <sup>18</sup>F-rhPSMA-7.3 (SAF)

| Descripted of Planned Arm | Subject<br>Identifier for<br>the Study | Visit<br>Name | Start Date/time (Study Day) | Planned Time Point<br>Name | Injection site reaction | Site of administration | Total Volume of undiluted IMP (mL) | Total administration activity (MBq) | Administration per protocol | Injection site reaction |
|---|---|---|---|---|---|---|---|---|---|---|
| Study Arm | Subject ID | VISIT X | YYYY-MM-<br>DDTHH:MM (XX) | Time Point | XXX | XXX | xxx | XXX | XXX | xxx |


CLINICAL TRIAL CONSULTANTS AB


Study Code: BED-PSMA-101 CTC Project No: 213-22-2018

Vital Signs

### LISTING 16.2.4.2. VITAL SIGNS – BMI, HEIGHT AND WEIGHT (SAF)

| Description of<br>Planned Arm | Subject Identifier for the Study | Visit Name | Planned Time Point<br>Name | Date/Time of<br>Measurements<br>(Study Day) | Height (cm) | Weight (kg) | Body Mass<br>Index (kg/m²) |
|---|---|---|---|---|---|---|---|
| Study Arm | Subject ID | VISIT X | Time point | YYYY-MM-DD<br>THH:MM (XX) | XXX | XX | XX.X |
| | ••• | | | ••• | | | |

### LISTING 16.2.4.3. VITAL SIGNS (SAF)

| Description of Planned Arm | Subject Identifier for the Study | Visit Name | Planned Time Point<br>Name | Date/Time of<br>Measurements<br>(Study Day) | Temperature (C | Systolic Blood °) Pressure (mmHg | | | Respiratory<br>Rate<br>(breaths/min) |
|---|---|---|---|---|---|---|---|---|---|
| Study Arm | Subject ID | VISIT X | Time point | YYYY-MM-DD<br>THH:MM (XX) | XX.X | xxx | XXX | XX | XX |
| ••• | ••• | | ••• | ••• | ••• | ••• | | | ••• |

BED-PSMA-101\_213-22-2018\_SAP\_v1.0\_30OCT2019


CLINICAL TRIAL CONSULTANTS AB


Study Code: BED-PSMA-101 CTC Project No: 213-22-2018

12-lead ECG Measurements

BED-PSMA-101\_213-22-2018\_SAP\_v1.0\_30OCT2019

### LISTING 16.2.9. 12-LEAD ECG MEASUREMENTS (SAF)

| Description of Planned Arm | Subject Identifier for the Study | Visit Name | Planned Time Point<br>Name | Date/Time of ECG<br>(Study Day) | QRS Duration<br>Aggregate (ms) | | QTcF Interval<br>Aggregate (ms) | PR Interval (ms) | ECG Mean Heart<br>Rate (beats/min) | Interpretation of ECG results |
|---|---|---|---|---|---|---|---|---|---|---|
| Study Arm | Subject ID | VISIT X | Time point | YYYY-MM-<br>DDTHH:MM (xx) | xx | XX | XX | xx | XX | Normal/Abnormal.<br>NCS/Abnormal, CS |

CLINICAL TRIAL CONSULTANTS AB


Study Code: BED-PSMA-101 CTC Project No: 213-22-2018

Safety Laboratory Results – Haematology

### LISTING 16.2.10.1. LABORATORY VALUES. HAEMATOLOGY (SAF)

| Description of<br>Planned Arm | Subject Identifier for the Study | Lab Test or Examination<br>Name | Visit Name | Planned Time<br>Point Name | Date/Time of Specimen<br>Collection (Study Day) | Character<br>Result/Findin<br>g in Std<br>Format | Standard<br>Units | Normal Range<br>Indicator | Lower<br>Reference<br>Limit | Upper<br>Reference<br>Limit | Interpretation |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Arm | Subject ID | Haemoglobin | VISIT X | Time point | YYYY-MM-<br>DDTHH:MM (XX) | XX | g/L | x | X | X | х |
| | | | | | | | | | ••• | ••• | |
| Study Arm | Subject ID | Haematocrit | VISIT X | Time point | YYYY-MM-<br>DDTHH:MM (XX) | XX | L/L | x | x | X | x |
| | | | | | | | | | ••• | | |
| Study Arm | Subject ID | Erythrocytes | VISIT X | Time point | YYYY-MM-<br>DDTHH:MM (XX) | xx | 10^12/L | x | x | X | x |
| Study Arm | Subject ID | MCV | VISIT X | Time point | YYYY-MM-<br>DDTHH:MM (XX) | XX | | X | x | X | x |
| Study Arm | Subject ID | MCH | VISIT X | Time point | YYYY-MM-<br>DDTHH:MM (XX) | xx | pg/cell | x | X | X | X |
| ••• | | | ••• | ••• | | | | | | | ••• |
| Study Arm | Subject ID | Platelets | VISIT X | Time point | YYYY-MM-<br>DDTHH:MM (XX) | XX | 10^9/L | x | X | X | x |
| ••• | | | | | | | | ••• | | | |
| Study Arm | Subject ID | Neutrophils | VISIT X | Time point | YYYY-MM-<br>DDTHH:MM (XX) | XX | 10^9/L | X | x | X | x |
| | | | ••• | | | ••• | ••• | ••• | ••• | ••• | |





| Description of Planned Arm | Subject Identifier for the Study | Lab Test or Examination<br>Name | Visit Name | Planned Time<br>Point Name | Date/Time of Specimen<br>Collection (Study Day) | Character<br>Result/Findin<br>g in Std<br>Format | Standard<br>Units | Normal Range<br>Indicator | Lower<br>e Reference<br>Limit | Upper<br>Reference<br>Limit | Interpretation |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Arm | Subject ID | Eosinophils | VISIT X | Time point | YYYY-MM-<br>DDTHH:MM (XX) | XX | 10^9/L | х | х | X | X |
| Study Arm | Subject ID | Basophils | VISIT X | Time point | YYYY-MM-<br>DDTHH:MM (XX) | xx | 10^9/L | X | X | X | X |
| | | | | | ••• | | ••• | | ••• | | |
| Study Arm | Subject ID | Lymphocytes | VISIT X | Time point | YYYY-MM-<br>DDTHH:MM (XX) | xx | 10^9/L | X | X | x | X |
| | | | ••• | | ••• | | ••• | | | ••• | |
| Study Arm | Subject ID | Monocytes | VISIT X | Time point | YYYY-MM-<br>DDTHH:MM (XX) | XX | 10^9/L | X | х | x | X |


Study Code: BED-PSMA-101 CTC Project No: 213-22-2018



Safety Laboratory Results – Clinical Chemistry

### LISTING 16.2.10.2. LABORATORY VALUES – CLINICAL CHEMISTRY (SAF)

| Description of<br>Planned Arm | Subject Identifier for the Study | Lab Test or Examination Name | Visit Name | Planned Time Point<br>Name | Date/Time of Specimen<br>Collection (Study Day) | Character<br>Result/Finding<br>in Std Format | Standard<br>Units | Normal<br>Range<br>Indicator | Lower<br>Reference<br>Limit | Upper<br>Reference<br>Limit | Interpretation |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Arm | Subject ID | Alkaline phosphatase | VISIT X | Time point | YYYY-MM-DDTHH:MM (XX) | xx | U/L | x | x | х | х |
| | | | | | ••• | | | | | | |
| Study Arm | Subject ID | Alanine Aminotransferase | VISIT X | Time point | YYYY-MM-DDTHH:MM (XX) | xx | U/L | x | X | x | X |
| | | | | | ••• | | | | | | ••• |
| Study Arm | Subject ID | Aspartate aminotransferase | VISIT X | Time point | YYYY-MM-DDTHH:MM (XX) | XX | U/L | X | x | x | X |
| | | | | | ••• | | | | | | |
| Study Arm | Subject ID | Gamma-glutamyl transferase | VISIT X | Time point | YYYY-MM-DDTHH:MM (XX) | XX | U/L | X | x | x | X |
| | | | ••• | | | ••• | | | | | ••• |
| Study Arm | Subject ID | Albumin | VISIT X | Time point | YYYY-MM-DDTHH:MM (XX) | XX | g/L | x | X | X | X |
| | | | | | | | | | | | ••• |
| Study Arm | Subject ID | Total protein | VISIT X | Time point | YYYY-MM-DDTHH:MM (XX) | XX | unit | x | X | X | X |
| Study Arm | Subject ID | Total bilirubin | VISIT X | Time point | YYYY-MM-DDTHH:MM (XX) | xx | umol/L | x | x | x | X |
| | | | | | | | | | ••• | | ••• |
| Study Arm | Subject ID | Conjugated bilirubin | VISIT X | Time point | YYYY-MM-DDTHH:MM (XX) | XX | umol/L | x | X | X | X |
| | | | | | ••• | ••• | | | | | |
| Study Arm | Subject ID | Creatine | VISIT x | Time point | YYYY-MM-DDTHH:MM (XX) | XX | umol/L | x | X | X | X |
| | | | | | | | | | | | ••• |
| Study Arm | Subject ID | Blood Urea Nitrogen (BUN) | VISIT x | | YYYY-MM-DDTHH:MM (XX) | | mmol/L | | x | x | X |
| , | , | 25. ( - 1) | | 1 | , ( ) | | | | | | |





| Description of Planned Arm | Subject Identifier for the Study | Lab Test or Examination Name | Visit Name | Planned Time Point<br>Name | Date/Time of Specimen<br>Collection (Study Day) | Character<br>Result/Finding<br>in Std Format | Standard<br>Units | Normal<br>Range<br>Indicator | Lower<br>Reference<br>Limit | Upper<br>Reference<br>Limit | Interpretation |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | ••• | | | ••• | ••• | ••• | ••• | ••• | ••• |
| Study Arm | Subject ID | Chloride | VISIT x | Time point | YYYY-MM-DDTHH:MM (XX) | xx | mmol/L | x | X | x | X |
| | | | | | | | ••• | | | | |
| Study Arm | Subject ID | Potassium | VISIT x | Time point | YYYY-MM-DDTHH:MM (XX) | xx | mmol/L | | X | X | X |
| | | | | | | ••• | ••• | | ••• | ••• | ••• |
| Study Arm | Subject ID | Sodium | VISIT x | Time point | YYYY-MM-DDTHH:MM (XX) | XX | mmol/L | | X | X | X |
| Study Arm | Subject ID | C-reactive Protein | VISIT x | Time point | YYYY-MM-DDTHH:MM (XX) | XX | umol/L | | X | X | X |
| Study Arm | Subject ID | FSH (female volunteers only) | VISIT x | Time point | YYYY-MM-DDTHH:MM (XX) | XX | unit | | X | X | X |
| Study Arm | Subject ID | Serum β-hCG pregnancy test (female volunteers only) | VISIT x | Time point | YYYY-MM-DDTHH:MM (XX) | XX | unit | | X | x | X |


**CLINICAL TRIAL CONSULTANTS AB** 


CTC Project No: 213-22-2018

Safety Laboratory Results – Coagulation

### LISTING 16.2.10.3. LABORATORY VALUES - COAGULATION (SAF)

| Description of Planned Arm | Subject Identifier for the Study | Lab Test or Examination Name | Visit Name | Planned Time Point<br>Name | Specimen Collection (Study Day) | Character<br>Result/Finding<br>in Std Format | _ | s Interpretation |
|---|---|---|---|---|---|---|---|---|
| Study Arm | Subject ID | Activated Partial Thromboplastin Time | VISIT X | Time point | YYYY-MM-<br>DDTHH:MM<br>(XX) | XX | X | х |
| ••• | | | | ••• | | | ••• | |
| Study Arm | Subject ID | Prothrombin Intl. Normalized Ratio | VISIT X | Time point | YYYY-MM-<br>DDTHH:MM (xx) | XX | X | X |
| ••• | ••• | | | | | | | |




Study Code: BED-PSMA-101 CTC Project No: 213-22-2018

Safety Laboratory Results – Urine

### LISTING 16.2.10.4. LABORATORY VALUES - URINE (SAF)

| Description of Planned Arm | Subject Identifier for the Study | Lab Test or Examination Name | Visit Name | Planned Time Point | Date/Time of Specimen<br>Collection (study day) | Character<br>Result/Finding<br>in Std Format | | s Interpretation |
|---|---|---|---|---|---|---|---|---|
| Study Arm | Subject ID | рН | VISIT X | Time point | YYYY-MM-DDTHH:MM<br>(XX) | XX | XX | XX |
| | | | | | | ••• | | |
| Study Arm | Subject ID | RBC | VISIT X | Time point | YYYY-MM-DDTHH:MM<br>(XX) | xx | XX | XX |
| | | | ••• | | | | | ••• |
| Study Arm | Subject ID | WBC | VISIT X | Time point | YYYY-MM-DDTHH:MM<br>(XX) | XX | XX | XX |
| | | | | | | ••• | | |
| Study Arm | Subject ID | Nitrite | VISIT X | Time point | YYYY-MM-DDTHH:MM<br>(XX) | XX | XX | XX |
| | | | | | | | ••• | |
| Study Arm | Subject ID | Protein | VISIT X | Time point | YYYY-MM-DDTHH:MM<br>(XX) | XX | XX | XX |
| | | | | | | ••• | ••• | |
| Study Arm | Subject ID | Glucose | VISIT X | Time point | YYYY-MM-DDTHH:MM<br>(XX) | XX | XX | XX |
| | | | | | | ••• | ••• | |
| Study Arm | Subject ID | Ketones | VISIT X | Time point | YYYY-MM-DDTHH:MM<br>(XX) | XX | xx | XX |
| | | | | ••• | | ••• | ••• | ••• |


CLINICAL TRIAL CONSULTANTS AB


CTC Project No: 213-22-2018

# **Physical Examinations**

### LISTING 16.2.11. PHYSICAL EXAMINATIONS (SAF)

| Subject<br>Identifier for | | Date/Time of Examination | | Eyes, Ears,<br>Nose, | | | | | | Peripheral | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| the Study | Visit name | (Study Day) | Abdominal | Cardiac | Dermatologic | Throat | Head | Lymphati | c Musculoskeletal | Neurologic | Vascular | Pulmonary |
| Subject ID | VISIT X | YYYY-MM-<br>DDTHH:MM<br>(xx) | XXX | XXX | XXX | XXX | xxx | XXX | xxx | XXX | xxx | xxx |





CTC Project No: 213-22-2018

Gleason Grade and Score

### LISTING 16.2.12. GLEASON GRADE AND SCORE (SAF)

| Subject<br>Identifier for<br>the Study | Date/Time of Test | Study Day | Primary Grade | Secondary Grade | Tertiary Grade | Gleason Grade |
|---|---|---|---|---|---|---|
| Subject ID | YYYY-MM-DD | xx | xxx | xxx | xxx | xxx |
| Subject ID | YYYY-MM-DD | xx | xxx | xxx | xxx | xxx |
| Subject ID | YYYY-MM-DD | xx | xxx | xxx | xxx | xxx |
| Subject ID | YYYY-MM-DD | xx | xxx | XXX | XXX | XXX |
| | | | | | | ••• |


CTC Project No: 213-22-2018

Histopathology Results



LISTING 16.2.13. HISTOPATHOLOGY RESULTS (SAF)


CLINICAL TRIAL CONSULTANTS AB


Study Code: BED-PSMA-101 CTC Project No: 213-22-2018

Adverse Events

#### LISTING 16.2.14.1. ADVERSE EVENTS PART 1 (ALL SUBJECTS)

| Description of Planned Arm | Subject<br>Identifier for<br>the Study | Reported Term for the Adverse<br>Event | Serious<br>Event | Start Date/Time of<br>Adverse Event<br>(Study Day) | End Date/Time of<br>Adverse Event<br>(Study Day) | Action Taken with Study<br>Treatment | Outcome of Adverse Event | Description of Element |
|---|---|---|---|---|---|---|---|---|
| Study Arm | Subject ID | Reported Term | Y/N | YYYY-MM-DD<br>THH:MM (xx) | YYYY-MM-DD<br>THH:MM (xx) | Action | Outcome | Treatment<br>Element |
| | | ••• | | | | | | |

#### LISTING 16.2.14.2. ADVERSE EVENTS PART 2 (ALL SUBJECTS)

| Description of Planned Arm | Subject Identifier for the Study | Reported<br>Term/Preferred<br>term/System organ<br>class | Start<br>date/time/Study day | End date/time (Study day) | Treatment emergent | Severity/intensity | Causality | Action | Outcome |
|---|---|---|---|---|---|---|---|---|---|
| Study Arm | Subject ID | Reported<br>term/AEDECOD/AEB<br>ODSYS | YYYY-MM-<br>DDTHH:MM/xxx | YYYY-MM-<br>DDTHH:MM<br>(xx) | Y/N | MILD/MODERATE/<br>SEVERE | RELATED/UNRELATED | xxx | xxx |
| ••• | ••• | ••• | ••• | ••• | | ••• | ••• | | ••• |


CLINICAL TRIAL CONSULTANTS AB


Study Code: BED-PSMA-101 CTC Project No: 213-22-2018

Serious Adverse Events

### LISTING 16.2.15.1. SERIOUS ADVERSE EVENTS PART 1 (ALL SUBJECTS)

| Description of<br>Planned Arm | Subject Identifier for the Study | Sequence<br>Number | Reported Term for the Adverse<br>Event | Serious<br>Event | Start Date/Time of<br>Adverse Event<br>(Study Day) | End Date/Time of<br>Adverse Event<br>(Study Day) | Action Taken with Study<br>Treatment | Outcome of Adverse Event | Description of Element |
|---|---|---|---|---|---|---|---|---|---|
| Study Arm | Subjects ID | X | Reported Term | Y/N | YYYY-MM-DD<br>THH:MM (xx) | YYYY-MM-DD<br>THH:MM (xx) | Action | Outcome | Treatment Group |
| | | | LISTING 16.2.15.2. S | SERIOUS . | ADVERSE EVENT | S PART 2 (ALL SUI | BJECTS) | | |
| Description of<br>Planned Arm | Subject Identifier for the Study | Sequence<br>Number | Reported Term for the Adverse<br>Event | Serious<br>Event | Dictionary-<br>Derived Term | Body System or<br>Organ Class | Severity/intensity | Causality | Description of Element |
| Study Arm | Subject ID | х | Reported Term | Y/N | Term | xxx | MILD/MODERATE/SE<br>VERE | RELATED/UNRELATED | xxx |
| | | | LISTING 16.2.15.3. SERIOUS A | ADVERSE | EVENTS – SERIO | USNESS CRITERIA | A (ALL SUBJECTS) | | |
| Description of Planned Arm | Subject Identifier for the Study | Sequence<br>Number | Reported Term for the Adverse<br>Event | Serious<br>Event | Start Date/Time of<br>Adverse Event<br>(Study Day) | End Date/Time of<br>Adverse Event<br>(Study Day) | Action Taken with Study<br>Treatment | Outcome of Adverse Event | Description of Element |
| Study Arm | Subject ID | Х | Action | Y/N | YYYY-MM-DD<br>THH:MM (xx) | YYYY-MM-DD<br>THH:MM (xx) | Action | Outcome | Treatment Group |
